CLINICAL TRIAL: NCT00550446
Title: A Phase 2b, Randomized, Double Blind, Placebo Controlled Active Comparator, Multicenter Study To Compare 5 Dose Regimens Of CP- 690,550 And Adalimumab Versus Placebo, Administered For 6 Months In The Treatment Of Subjects With Active Rheumatoid Arthritis
Brief Title: A Phase 2 Study For Patients With A Physician's Diagnosis Of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921035
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Janus Kinase 3 Clinical Trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Active Comparator)
  Interventions: Drug: Adalimumab
- 2 (Experimental)
  Interventions: Drug: CP-690-550
- 3 (Experimental)
  Interventions: Drug: CP-690-550
- 4 (Experimental)
  Interventions: Drug: CP-690-550
- 5 (Experimental)
  Interventions: Drug: CP-690,550
- 6 (Experimental)
  Interventions: Drug: CP-690,550
- 7 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — 40mg subcutaneous injections every other week for 6 injections during week 0-10 with oral placebo BID. Subjects switched to CP-690,550 at week 12.
  Arms: 1
Drug: CP-690-550 — 15 mg BID oral plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 2
Drug: CP-690-550 — 10 mg BID oral plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 3
Drug: CP-690-550 — 5 mg BID oral plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 4
Drug: CP-690,550 — 3 mg BID PO plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 5
Drug: CP-690,550 — 1 mg BID PO plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 6
Drug: Placebo — Placebo by mouth plus 6 placebo subcutaneous injections (week 0-10)
  Arms: 7

SUMMARY:
The purpose of this study is to determine the effectiveness and safety, over 6 months, of 5 doses of CP-690,550 for the treatment of adults with active rheumatoid arthritis. Five out of seven subjects will receive CP-690,550. One out of seven will receive adalimumab (Humira®) and one out of seven will only receive inactive substances (placebo.)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have active rheumatoid arthritis
* Subjects must have failed at least 1 disease modifying anti-rheumatic drug (DMARD)
* Subjects must not be currently taking any DMARD other than an antimalarial

Exclusion Criteria:

* Subjects who discontinued any previous TNF inhibitor therapy for either lack of benefit or safety.
* Subjects who previously received adalimumab (Humira®) therapy for any reason.
* Subjects with evidence of blood disorders, chronic infections or untreated tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (20):
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Mesquite, Texas
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (2):
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Sofia
- Chile (2):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
- Croatia (2):
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Zagreb
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 11 - Chodov
  - Pfizer Investigational Site, Zlín
- Germany (4):
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hildesheim
  - Pfizer Investigational Site, Leipzig
- Greece (2):
  - Pfizer Investigational Site, Goudi, Athens
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Szolnok, Hungary
- Italy (2):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Genova
- Mexico (4):
  - Pfizer Investigational Site, México, D.f.
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Cuernavaca, Morelos
  - Pfizer Investigational Site, Metepec, State of Mexico
- Romania (3):
  - Pfizer Investigational Site, Constanța, Constanța County
  - Pfizer Investigational Site, Iași, Iaşi
  - Pfizer Investigational Site, Bucharest
- Slovakia (2):
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Žilina
- Pfizer Investigational Site, Seoul, South Korea
- Ukraine (5):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Vinnitsa
  - Pfizer Investigational Site, Zaporizhzhia

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Suzuki M, Shoji S, Miyoshi S, Krishnaswami S. Model-Based Comparison of Dose-Response Profiles of Tofacitinib in Japanese Versus Western Rheumatoid Arthritis Patients. J Clin Pharmacol. 2020 Feb;60(2):198-208. doi: 10.1002/jcph.1514. Epub 2019 Sep 12. PMID 31512746
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Wallenstein GV, Kanik KS, Wilkinson B, Cohen S, Cutolo M, Fleischmann RM, Genovese MC, Gomez Reino J, Gruben D, Kremer J, Krishnaswami S, Lee EB, Pascual-Ramos V, Strand V, Zwillich SH. Effects of the oral Janus kinase inhibitor tofacitinib on patient-reported outcomes in patients with active rheumatoid arthritis: results of two Phase 2 randomised controlled trials. Clin Exp Rheumatol. 2016 May-Jun;34(3):430-42. Epub 2016 Apr 28. PMID 27156561
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Fleischmann R, Cutolo M, Genovese MC, Lee EB, Kanik KS, Sadis S, Connell CA, Gruben D, Krishnaswami S, Wallenstein G, Wilkinson BE, Zwillich SH. Phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) or adalimumab monotherapy versus placebo in patients with active rheumatoid arthritis with an inadequate response to disease-modifying antirheumatic drugs. Arthritis Rheum. 2012 Mar;64(3):617-29. doi: 10.1002/art.33383. PMID 21952978
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921035&StudyName=A%20Phase%202%20Study%20For%20Patients%20With%20A%20Physician%27s%20Diagnosis%20Of%20Rheumatoid%20Arthritis%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 1 mg: CP-690,550 1 milligram (mg) tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10. Participants who failed to achieve a minimum improvement of at least 20 percent (%) reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 1 mg to 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 3 mg: CP-690,550 3 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 3 mg to 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.
- CP-690,550 15 mg: CP-690,550 15 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.
- Adalimumab: Adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10 along with placebo matched to CP-690,550 tablet orally twice daily up to Week 12, then CP-690,550 5 mg tablet orally twice daily up to Week 24.
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections QOW up to Week 10. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to placebo to 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 1 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 1 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- CP-690,550 3 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 3 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- Adalimumab to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in adalimumab 40 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- Placebo to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in placebo treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
Period: Up To Week 12
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Placebo | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg to CP-690,550 5 mg (R) | Adalimumab to CP-690,550 5 mg (R) | Placebo to CP-690,550 5 mg (R)
Started | 54 | 52 | 50 | 61 | 57 | 53 | 59 | 0 | 0 | 0 | 0
Treated | 54 | 51 | 49 | 61 | 57 | 53 | 59 | 0 | 0 | 0 | 0
Completed | 44 | 47 | 46 | 58 | 54 | 45 | 46 | 0 | 0 | 0 | 0
Not Completed | 10 | 5 | 4 | 3 | 3 | 8 | 13 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Randomized not treated | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post Week 12
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Placebo | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg to CP-690,550 5 mg (R) | Adalimumab to CP-690,550 5 mg (R) | Placebo to CP-690,550 5 mg (R)
Started | 27 | 30 | 46 | 58 | 54 | 1 | 21 | 17 | 17 | 44 | 25
Completed | 24 | 28 | 43 | 55 | 52 | 0 | 19 | 16 | 15 | 37 | 24
Not Completed | 3 | 2 | 3 | 3 | 2 | 1 | 2 | 1 | 2 | 7 | 1
Not completed — Adverse Event | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 1 mg: CP-690,550 1 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 1 mg to 5 mg (R) treatment arm for next 12 weeks.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Placebo | Total
Number analyzed (Participants) | 54 | 51 | 49 | 61 | 57 | 53 | 59 | 384
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.3) | 53.4 (12.2) | 53.7 (13.5) | 52.4 (10.9) | 53.2 (13.0) | 53.5 (11.9) | 52.5 (13.7) | 53.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 43 | 53 | 50 | 45 | 52 | 333
  Male | 8 | 7 | 6 | 8 | 7 | 8 | 7 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: greater than or equal to (>=) 20 % improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. The analysis used Baseline Observation Carried Forward (BOCF) imputation for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Placebo
Number analyzed (Participants) | 54 | 51 | 49 | 61 | 57 | 53 | 59
percentage of participants | 31.48 | 45.10 | 61.22 | 72.13 | 71.93 | 39.62 | 23.73

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: 20% improvement in TJC; >=20% improvement in SJC; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 10, 16, 20 and 24/Early Termination (ET)
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Missing values were imputed using BOCF. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
percentage of participants
  Week 2 (n=54,0,51,0,49,61,57,53,0,59,0) | 16.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.37 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.65 | 50.82 | 38.60 | 26.42 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=54,0,51,0,49,61,57,53,0,59,0) | 22.22 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.82 | 52.46 | 63.16 | 28.30 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.12 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=54,0,51,0,49,61,57,53,0,59,0) | 38.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.06 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 63.27 | 63.93 | 66.67 | 30.19 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 25.42 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=54,0,51,0,49,61,57,53,0,59,0) | 37.04 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.06 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 63.27 | 65.57 | 71.93 | 35.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.12 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=54,0,51,0,49,61,57,53,0,59,0) | 35.19 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 57.14 | 75.41 | 75.44 | 35.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 23.73 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=37,17,34,17,49,61,57,9,44,34,25) | 51.4 | 0.0 | 58.8 | 0.0 | 67.3 | 70.5 | 71.9 | 0.0 | 0.0 | 35.3 | 0.0
  Week 20 (n=37,17,34,17,49,61,57,9,44,34,25) | 45.9 | 0.0 | 64.7 | 0.0 | 69.4 | 73.8 | 71.9 | 0.0 | 0.0 | 32.4 | 0.0
  Week 24 (n=37,17,34,17,49,61,57,9,44,34,25) | 35.1 | 0.0 | 58.8 | 0.0 | 57.1 | 73.8 | 68.4 | 0.0 | 0.0 | 47.1 | 0.0

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50%(ACR50) Response
Description: ACR50 response: >= 50% improvement in TJC or SJC and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
percentage of participants
  Week 2 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.84 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.16 | 18.03 | 17.54 | 7.55 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=54,0,51,0,49,61,57,53,0,59,0) | 9.26 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.73 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.20 | 31.15 | 40.35 | 9.43 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.08 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=54,0,51,0,49,61,57,53,0,59,0) | 14.81 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.29 | 36.07 | 42.11 | 16.98 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.78 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=54,0,51,0,49,61,57,53,0,59,0) | 12.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.57 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.49 | 29.51 | 49.12 | 16.98 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.47 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=54,0,51,0,49,61,57,53,0,59,0) | 12.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.65 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.69 | 50.82 | 43.86 | 15.09 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.78 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=54,0,51,0,49,61,57,53,0,59,0) | 11.11 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 25.49 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.78 | 45.90 | 50.88 | 20.75 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.17 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=37,17,34,17,49,61,57,9,44,34,25) | 18.9 | 0.0 | 38.2 | 0.0 | 34.7 | 42.6 | 56.1 | 0.0 | 0.0 | 20.6 | 0.0
  Week 20 (n=37,17,34,17,49,61,57,9,44,34,25) | 18.9 | 0.0 | 44.1 | 0.0 | 32.7 | 42.6 | 59.6 | 0.0 | 0.0 | 17.6 | 0.0
  Week 24 (n=37,17,34,17,49,61,57,9,44,34,25) | 10.8 | 0.0 | 44.1 | 0.0 | 36.7 | 45.9 | 54.4 | 0.0 | 0.0 | 17.6 | 0.0

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >= 70% improvement in TJC or SJC and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Missing values were imputed using BOCF. n=number of participants evaluable at specific time points for each arm group respectively.
Measure: Number; unit: percentage of participants
Groups:
- CP-690,550 15 mg: CP-690,550 15 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.CP-690,550 15 mg tablet orally twice daily plus placebo QOW subcutaneous injections during Week 0 to Week 10.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
percentage of participants
  Week 2 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.04 | 3.28 | 7.02 | 1.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=54,0,51,0,49,61,57,53,0,59,0) | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.88 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.04 | 11.48 | 8.77 | 5.66 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=54,0,51,0,49,61,57,53,0,59,0) | 3.70 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.08 | 19.67 | 17.54 | 5.66 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=54,0,51,0,49,61,57,53,0,59,0) | 9.26 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.92 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.16 | 18.03 | 24.56 | 5.66 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=54,0,51,0,49,61,57,53,0,59,0) | 3.70 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.84 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.33 | 26.23 | 21.05 | 3.77 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.69 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=54,0,51,0,49,61,57,53,0,59,0) | 5.56 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.76 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.29 | 24.59 | 26.32 | 3.77 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.39 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=37,17,34,17,49,61,57,9,44,34,25) | 10.8 | 0.0 | 26.5 | 0.0 | 20.4 | 29.5 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0
  Week 20 (n=37,17,34,17,49,61,57,9,44,34,25) | 10.8 | 0.0 | 17.6 | 0.0 | 18.4 | 31.1 | 31.6 | 0.0 | 0.0 | 8.8 | 0.0
  Week 24 (n=37,17,34,17,49,61,57,9,44,34,25) | 8.1 | 0.0 | 23.5 | 0.0 | 22.4 | 37.7 | 33.3 | 0.0 | 0.0 | 11.8 | 0.0

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 90% (ACR90) Response
Description: ACR90 response: >= 90% improvement in TJC or SJC and 90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
percentage of participants
  Week 2 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | 1.64 | 0.00 | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=54,0,51,0,49,61,57,53,0,59,0) | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.04 | 3.28 | 1.75 | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=54,0,51,0,49,61,57,53,0,59,0) | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.04 | 6.56 | 1.75 | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.04 | 9.84 | 1.75 | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.08 | 9.84 | 10.53 | 1.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=54,0,51,0,49,61,57,53,0,59,0) | 1.85 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.96 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.08 | 11.48 | 7.02 | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=37,17,34,17,49,61,57,9,44,34,25) | 2.7 | 0.0 | 5.9 | 0.0 | 8.2 | 13.1 | 8.8 | 0.0 | 0.0 | 0.0 | 0.0
  Week 20 (n=37,17,34,17,49,61,57,9,44,34,25) | 2.7 | 0.0 | 2.9 | 0.0 | 6.1 | 11.5 | 10.5 | 0.0 | 0.0 | 0.0 | 0.0
  Week 24 (n=37,17,34,17,49,61,57,9,44,34,25) | 2.7 | 0.0 | 5.9 | 0.0 | 6.1 | 14.8 | 12.3 | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Area Under the Numeric Index of American College of Rheumatology Response (ACR-n) Curve
Description: ACR-n = calculated for each participant by taking the lowest percentage improvement in (1) SJC or (2) TJC or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening. Area under the curve (AUC) for ACR-n is the measure of the area under the curve of the mean change from baseline in ACR-n. The trapezoidal rule was used to compute the AUC.
Time Frame: Baseline up to Week 2, 4, 6, 8, 10, 12
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure. Missing values were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Placebo
Number analyzed (Participants) | 54 | 50 | 49 | 61 | 56 | 53 | 59
units on a scale
  Week 2 | -99.17 (430.60) | -21.41 (348.60) | 36.11 (254.60) | 117.91 (236.40) | 16.24 (507.70) | -82.12 (436.48) | -97.56 (362.62)
  Week 4 | -328.58 (1190.65) | -31.17 (1068.34) | 165.07 (685.88) | 421.90 (700.43) | 184.76 (1317.14) | -211.66 (1178.51) | -268.25 (906.61)
  Week 6 | -488.95 (2121.82) | -7.91 (1840.80) | 416.04 (1117.60) | 839.12 (1219.16) | 584.69 (1864.04) | -280.67 (1925.43) | -430.41 (1471.10)
  Week 8 | -545.16 (3121.09) | 30.98 (2675.04) | 761.40 (1552.54) | 1311.99 (1736.67) | 1077.41 (2543.43) | -331.79 (2727.74) | -531.80 (2095.50)
  Week 10 | -588.77 (4109.74) | 81.85 (3510.17) | 1163.37 (1985.69) | 1857.57 (2203.00) | 1539.51 (3768.28) | -337.47 (3478.31) | -642.56 (2805.90)
  Week 12 | -675.05 (5160.91) | 145.08 (4380.78) | 1579.56 (2447.05) | 2443.62 (2701.93) | 2053.03 (4745.53) | -242.83 (4111.62) | -803.67 (3548.72)

7. Secondary Outcome: Tender Joint Count (TJC)
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Groups:
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.CP-690,550 5 mg tablet orally twice daily plus placebo QOW subcutaneous injections during Week 0 to Week 10.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
tender joints
  Baseline (n=54,0,51,0,49,61,57,53,0,59,0) | 27.02 (15.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.55 (11.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.14 (14.62) | 25.70 (13.92) | 25.88 (13.37) | 24.11 (13.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 25.92 (12.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,48,60,57,53,0,57,0) | 21.98 (14.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.94 (10.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.79 (12.42) | 15.33 (12.74) | 17.42 (14.33) | 19.40 (14.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.00 (11.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | 20.54 (17.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.83 (11.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.43 (13.01) | 12.84 (12.55) | 13.16 (14.95) | 16.78 (14.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.94 (13.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | 15.13 (13.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.67 (12.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.33 (11.06) | 10.95 (11.95) | 11.27 (14.89) | 15.73 (13.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.77 (14.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | 16.30 (14.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.40 (12.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.68 (12.57) | 10.00 (11.81) | 9.15 (12.18) | 14.87 (13.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.93 (12.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 17.15 (17.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.65 (11.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.87 (11.17) | 7.68 (10.94) | 9.23 (12.88) | 14.47 (15.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.22 (14.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | 18.32 (16.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.33 (12.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.52 (12.35) | 8.09 (12.02) | 8.44 (11.26) | 14.74 (14.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.50 (13.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | 7.44 (8.38) | 19.47 (14.06) | 6.27 (6.49) | 19.41 (12.25) | 10.85 (11.11) | 7.57 (11.08) | 7.22 (11.34) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 8.70 (9.47) | 8.30 (9.07) | 12.40 (12.24)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | 10.41 (10.69) | 16.19 (9.72) | 6.76 (8.25) | 18.25 (15.65) | 11.80 (12.82) | 6.66 (10.62) | 6.79 (9.69) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 8.95 (10.56) | 8.16 (8.74) | 12.60 (13.28)
  Week 24 (n=24,16,29,15,43,55,52,0,39,20,24) | 11.92 (13.64) | 21.31 (14.81) | 6.59 (10.58) | 16.60 (13.49) | 10.47 (11.50) | 6.25 (10.12) | 7.27 (11.35) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 10.44 (9.97) | 8.75 (8.59) | 10.54 (13.09)

8. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24 or ET
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicated an improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 60 | 57 | 53 | 44 | 57 | 25
tender joints
  Week 2 (n=54,0,51,0,48,60,57,53,0,57,0) | -5.04 (12.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.61 (9.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.23 (12.61) | -10.28 (12.57) | -8.46 (12.87) | -4.72 (10.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.19 (11.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | -6.56 (14.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.43 (10.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.33 (10.76) | -13.00 (12.73) | -12.85 (14.91) | -7.67 (11.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.23 (11.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | -11.96 (15.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.38 (11.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.40 (13.50) | -14.49 (13.52) | -14.38 (14.86) | -8.83 (13.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.69 (13.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | -11.83 (13.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.65 (11.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.70 (13.86) | -15.61 (13.82) | -15.57 (13.80) | -8.57 (12.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.67 (11.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | -11.07 (16.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.65 (10.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.93 (13.92) | -17.51 (14.08) | -15.77 (12.77) | -9.89 (12.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.72 (13.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | -9.57 (15.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.04 (11.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.24 (13.32) | -16.74 (14.23) | -16.28 (12.25) | -9.30 (11.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.43 (14.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | -19.11 (13.88) | -10.53 (12.43) | -15.03 (9.88) | -8.47 (12.51) | -16.91 (13.06) | -17.48 (13.24) | -17.50 (13.29) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -15.09 (12.35) | -19.55 (13.02) | -12.40 (10.17)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | -16.15 (16.26) | -13.38 (11.59) | -15.28 (11.11) | -10.00 (13.23) | -15.98 (13.20) | -17.53 (12.86) | -17.57 (13.62) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -15.18 (11.25) | -18.16 (13.00) | -12.20 (12.02)
  Week 24 (n=24,16,29,15,43,55,52,0,39,20,24) | -12.63 (14.37) | -8.25 (13.75) | -15.45 (13.03) | -10.47 (13.60) | -17.58 (15.22) | -18.42 (13.64) | -17.02 (14.14) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -13.10 (12.94) | -19.10 (14.88) | -14.21 (12.25)

9. Secondary Outcome: Swollen Joint Counts (SJC)
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
swollen joints
  Baseline (n=54,0,51,0,49,61,57,53,0,59,0) | 16.70 (8.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.90 (8.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.35 (10.26) | 16.33 (8.28) | 16.93 (9.03) | 14.91 (8.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.90 (9.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,48,60,57,53,0,57,0) | 11.87 (7.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.82 (10.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.27 (8.90) | 10.55 (9.13) | 11.25 (8.91) | 11.58 (9.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.25 (8.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | 12.78 (13.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.98 (10.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.43 (9.15) | 8.50 (7.60) | 7.55 (8.89) | 10.08 (8.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.11 (9.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | 9.58 (9.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.08 (9.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.29 (5.77) | 7.03 (7.24) | 6.55 (8.02) | 9.27 (9.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.44 (11.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | 11.11 (11.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.88 (10.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.15 (7.46) | 7.02 (8.63) | 5.91 (7.65) | 8.89 (10.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.37 (9.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 10.63 (10.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.35 (9.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.93 (7.11) | 5.39 (7.47) | 5.68 (7.96) | 9.11 (11.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.76 (11.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | 11.39 (11.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.26 (10.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.33 (7.15) | 5.58 (7.84) | 5.11 (7.15) | 7.41 (7.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.85 (9.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | 6.44 (7.29) | 10.82 (7.63) | 4.50 (5.48) | 14.88 (13.15) | 5.96 (6.54) | 5.34 (7.91) | 4.46 (7.64) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 4.56 (5.59) | 5.90 (6.02) | 9.76 (8.53)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | 7.89 (7.95) | 10.31 (8.55) | 5.03 (7.59) | 14.38 (13.99) | 6.71 (6.96) | 4.60 (7.82) | 4.36 (7.17) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.52 (7.68) | 5.21 (4.50) | 7.92 (6.95)
  Week 24 (n=24,16,29,15,43,55,52,0,39,20,24) | 8.92 (11.01) | 10.94 (9.04) | 4.86 (7.81) | 13.27 (13.01) | 5.88 (6.38) | 4.44 (7.78) | 4.10 (6.83) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.67 (7.46) | 5.95 (6.26) | 6.04 (6.40)

10. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling = 1. A negative value in change from baseline indicated an improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: swollen joints
Groups:
- CP-690,550 3 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 3 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.Initially CP-690,550 3 mg tablet administered orally twice daily plus placebo QOW subcutaneous injections during Week 0 to Week 10. After Week 12, participants were reassigned CP-690,550 5 mg tablet administered orally twice daily.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Week 24, along with placebo matched to adalimumab 40 mg subcutaneous injections every other week (QOW) up to Week 10.CP-690,550 10 mg tablet orally twice daily plus placebo QOW subcutaneous injections during Week 0 to Week 10.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 60 | 57 | 53 | 44 | 57 | 25
swollen joints
  Week 2 (n=54,0,51,0,48,60,57,53,0,57,0) | -4.83 (7.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.08 (8.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.85 (9.65) | -5.67 (6.94) | -5.68 (9.98) | -3.32 (9.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.74 (8.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | -4.08 (10.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.66 (9.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.63 (9.01) | -8.02 (7.03) | -9.55 (11.00) | -4.57 (8.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.06 (8.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | -7.88 (9.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.54 (9.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.69 (9.13) | -9.36 (7.60) | -10.51 (10.61) | -5.75 (8.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.87 (10.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | -6.36 (10.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.75 (9.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.70 (9.60) | -9.19 (7.70) | -10.85 (10.60) | -6.17 (8.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.33 (9.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | -6.70 (8.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.33 (9.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.89 (9.78) | -11.11 (7.99) | -11.28 (10.79) | -6.00 (9.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.50 (11.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | -6.07 (9.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.85 (10.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.74 (10.28) | -10.91 (8.48) | -11.65 (10.26) | -7.83 (7.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.41 (9.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | -11.00 (8.75) | -6.65 (9.84) | -9.97 (6.98) | -1.24 (13.15) | -11.11 (9.87) | -11.27 (8.86) | -12.30 (10.98) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -10.86 (8.03) | -10.25 (6.77) | -7.00 (11.08)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | -9.56 (9.21) | -6.06 (9.70) | -9.90 (9.32) | -2.19 (14.28) | -10.40 (10.40) | -11.17 (7.92) | -12.68 (10.65) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -9.91 (7.50) | -11.47 (7.46) | -8.84 (9.92)
  Week 24 (n=24,16,29,15,43,55,52,0,39,20,24) | -8.58 (8.98) | -5.44 (9.33) | -10.07 (9.70) | -1.60 (14.34) | -11.60 (11.55) | -11.75 (7.82) | -13.10 (10.44) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -9.46 (9.37) | -10.20 (7.78) | -11.00 (11.16)

11. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
mm
  Baseline (n=54,0,51,0,49,61,56,53,0,59,0) | 59.74 (23.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 61.25 (23.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 64.14 (23.55) | 62.92 (18.74) | 63.46 (25.26) | 64.36 (21.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 60.29 (23.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,48,60,57,53,0,57,0) | 53.76 (24.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.25 (24.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.10 (24.48) | 43.90 (23.43) | 41.28 (28.06) | 48.00 (25.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 55.26 (26.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | 51.72 (24.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.91 (23.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.65 (22.56) | 33.28 (22.37) | 32.69 (23.77) | 46.78 (23.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.89 (23.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | 47.31 (24.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.75 (22.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.24 (22.73) | 33.68 (22.52) | 30.24 (25.46) | 46.27 (28.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.63 (24.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | 47.28 (25.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.21 (22.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.91 (23.56) | 33.05 (22.34) | 26.74 (26.01) | 43.17 (25.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.26 (23.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 45.70 (26.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.24 (23.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.67 (24.34) | 28.11 (21.80) | 23.38 (22.03) | 48.73 (27.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.96 (24.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | 47.25 (25.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.30 (26.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.70 (25.23) | 28.14 (22.79) | 27.26 (25.88) | 42.87 (25.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.93 (24.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | 35.00 (26.63) | 49.29 (29.81) | 34.97 (29.16) | 47.88 (25.87) | 31.39 (23.72) | 29.05 (26.23) | 24.24 (23.60) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 30.16 (21.52) | 37.55 (22.42) | 28.16 (22.28)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | 39.67 (27.28) | 43.38 (24.69) | 34.66 (29.75) | 38.81 (25.45) | 33.13 (24.57) | 27.43 (23.98) | 23.21 (22.60) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 31.68 (22.68) | 36.95 (25.80) | 31.64 (20.22)
  Week 24 (n=24,16,29,15,43,55,52,0,40,20,24) | 44.13 (24.32) | 44.00 (28.63) | 30.62 (28.36) | 31.87 (20.47) | 31.81 (27.72) | 22.85 (22.04) | 25.31 (22.28) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 34.33 (24.87) | 31.35 (22.51) | 29.83 (18.37)

12. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: as for outcome 11
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 60 | 56 | 53 | 44 | 57 | 25
mm
  Week 2 (n=54,0,51,0,48,60,56,53,0,57,0) | -5.98 (25.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.00 (17.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.33 (20.70) | -19.33 (22.50) | -23.11 (29.72) | -16.36 (23.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.14 (25.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,54,49,0,53,0) | -6.78 (30.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -19.04 (19.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -20.28 (21.33) | -28.60 (24.09) | -32.41 (29.39) | -16.96 (28.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.89 (23.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,54,48,0,52,0) | -11.42 (28.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.23 (23.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -25.04 (22.63) | -28.80 (22.13) | -33.50 (29.39) | -18.35 (26.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.08 (22.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | -11.68 (29.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -18.77 (20.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -30.02 (25.59) | -29.07 (23.84) | -35.83 (30.52) | -20.83 (27.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.28 (23.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | -13.98 (27.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.39 (22.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -29.30 (26.46) | -34.77 (25.60) | -38.94 (29.33) | -16.80 (26.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.63 (21.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | -11.61 (31.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.04 (22.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -31.24 (24.72) | -34.47 (25.63) | -35.31 (31.92) | -23.15 (27.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.65 (24.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | -19.00 (33.30) | -17.29 (29.71) | -18.73 (25.91) | -21.00 (22.29) | -32.54 (23.55) | -33.77 (27.27) | -38.33 (30.31) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -36.37 (22.95) | -16.05 (24.30) | -33.40 (25.97)
  Week 20 (n=27,16,29,16,45,53,53,0,44,19,25) | -14.33 (28.92) | -22.19 (29.73) | -19.66 (25.00) | -29.50 (25.80) | -31.67 (20.98) | -34.66 (23.72) | -39.55 (31.04) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -35.09 (27.62) | -15.58 (25.51) | -29.92 (23.24)
  Week 24 (n=24,16,29,15,43,55,52,0,40,20,24) | -9.83 (29.65) | -21.56 (35.86) | -23.69 (24.12) | -36.00 (18.57) | -32.84 (25.37) | -39.69 (22.62) | -37.83 (28.84) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -31.48 (28.90) | -22.25 (25.21) | -31.63 (24.22)

13. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 44 | 59 | 25
mm
  Baseline (n=54,0,51,0,49,61,57,53,0,59,0) | 60.74 (24.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 59.76 (22.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 67.55 (22.44) | 62.41 (19.94) | 62.77 (27.24) | 62.15 (21.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 61.41 (21.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=53,0,51,0,48,60,57,53,0,57,0) | 54.36 (23.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 48.49 (24.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.58 (24.55) | 41.82 (24.09) | 42.02 (25.77) | 48.00 (24.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 58.93 (25.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | 52.96 (23.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.68 (23.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.54 (23.10) | 34.86 (23.15) | 34.73 (25.05) | 46.24 (23.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.40 (23.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | 47.08 (23.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.52 (21.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.07 (22.47) | 33.63 (22.01) | 31.09 (25.20) | 43.46 (25.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.71 (22.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | 46.57 (27.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.02 (23.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.81 (23.95) | 33.42 (23.39) | 28.07 (26.86) | 43.85 (23.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.74 (23.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 45.80 (27.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.57 (24.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.04 (24.26) | 29.09 (21.52) | 22.72 (23.36) | 46.11 (25.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.24 (24.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | 45.39 (26.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.78 (26.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.52 (24.26) | 29.02 (23.09) | 26.39 (26.55) | 44.04 (25.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.85 (23.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | 36.07 (25.88) | 52.00 (28.93) | 35.03 (29.52) | 44.24 (25.78) | 30.37 (23.58) | 30.71 (25.69) | 24.72 (23.11) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 31.33 (18.80) | 38.65 (22.37) | 32.48 (20.69)
  Week 20 (n=27,16,29,16,45,53,52,0,44,19,25) | 39.74 (27.72) | 47.19 (24.36) | 35.41 (29.13) | 41.44 (24.86) | 33.91 (24.90) | 28.06 (23.26) | 23.90 (22.38) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 30.95 (21.47) | 35.84 (26.21) | 36.20 (21.44)
  Week 24 (n=24,16,29,15,43,55,52,0,40,20,24) | 43.08 (23.92) | 45.69 (26.15) | 33.07 (27.90) | 33.20 (19.77) | 33.77 (28.44) | 24.85 (22.29) | 26.58 (23.04) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 34.45 (23.60) | 32.05 (22.63) | 28.13 (17.42)

14. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) of Arthritis at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: as for outcome 13
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 53 | 17 | 51 | 17 | 48 | 60 | 57 | 53 | 44 | 57 | 25
mm
  Week 2 (n=53,0,51,0,48,60,57,53,0,57,0) | -5.72 (22.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.27 (18.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.33 (26.14) | -21.48 (25.18) | -20.75 (28.26) | -14.15 (25.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.84 (26.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | -6.62 (28.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.51 (22.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -23.15 (24.65) | -26.52 (25.06) | -28.29 (28.34) | -15.35 (25.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.64 (22.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,45,59,55,48,0,52,0) | -13.58 (29.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.77 (25.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -28.89 (24.62) | -28.39 (25.53) | -31.49 (29.39) | -18.69 (24.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.27 (18.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | -13.79 (27.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.27 (21.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -32.91 (28.68) | -28.18 (26.81) | -34.11 (29.33) | -18.23 (29.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.24 (19.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | -14.70 (26.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.21 (21.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -32.93 (28.11) | -33.21 (27.96) | -39.25 (28.87) | -17.42 (26.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.93 (22.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | -15.05 (29.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.96 (22.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -34.17 (25.62) | -33.09 (28.82) | -35.80 (30.90) | -19.80 (29.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.33 (22.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,54,0,43,20,25) | -19.81 (29.62) | -15.65 (29.98) | -20.60 (24.26) | -19.35 (22.34) | -37.33 (25.23) | -31.50 (28.85) | -37.46 (29.80) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -33.19 (25.10) | -16.75 (24.67) | -32.44 (22.40)
  Week 20 (n=27,16,29,16,45,53,52,0,44,19,25) | -16.15 (30.54) | -19.69 (31.12) | -20.38 (23.79) | -21.00 (17.74) | -34.73 (24.52) | -32.87 (24.10) | -37.65 (32.14) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -33.64 (28.30) | -18.74 (20.40) | -28.72 (22.80)
  Week 24 (n=24,16,29,15,43,55,52,0,40,20,24) | -12.96 (26.46) | -21.19 (33.96) | -22.72 (25.10) | -27.93 (15.08) | -34.72 (26.19) | -37.31 (25.58) | -36.10 (29.30) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -29.33 (34.25) | -23.35 (16.74) | -36.75 (21.95)

15. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis
Description: Physician global assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 60 | 57 | 53 | 44 | 57 | 25
mm
  Baseline (n=54,0,50,0,48,60,57,53,0,59,0) | 62.13 (16.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 62.10 (18.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 65.85 (14.36) | 61.05 (15.78) | 67.19 (17.93) | 62.77 (15.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 63.02 (18.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,46,60,57,53,0,57,0) | 52.30 (21.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.88 (20.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.37 (21.90) | 39.85 (18.69) | 44.98 (21.61) | 47.58 (20.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 55.19 (19.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,46,58,55,49,0,53,0) | 47.30 (20.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.23 (20.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.3 (19.49) | 34.55 (20.68) | 31.89 (20.38) | 44.02 (20.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.15 (20.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,47,0,45,59,55,48,0,52,0) | 39.75 (21.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.98 (21.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.40 (20.40) | 31.22 (19.51) | 28.56 (21.47) | 39.83 (22.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.12 (24.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,57,54,47,0,46,0) | 40.06 (22.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.54 (23.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.79 (19.94) | 29.56 (18.60) | 25.20 (21.85) | 38.34 (21.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.91 (20.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 41.65 (23.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.78 (24.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.70 (20.03) | 24.72 (18.83) | 23.68 (18.76) | 40.69 (25.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.83 (21.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,46,57,54,46,0,46,0) | 41.72 (23.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.65 (23.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.80 (19.13) | 25.37 (20.01) | 24.20 (18.74) | 38.22 (23.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.76 (24.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,56,53,0,43,20,25) | 29.93 (19.58) | 48.59 (20.92) | 26.97 (23.53) | 44.59 (21.99) | 29.74 (20.31) | 24.39 (19.14) | 21.09 (19.71) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 25.74 (15.96) | 28.70 (22.76) | 34.00 (20.65)
  Week 20 (n=27,16,29,16,45,52,53,0,44,19,25) | 32.59 (20.17) | 45.69 (15.98) | 23.86 (20.45) | 41.25 (23.77) | 27.04 (17.16) | 19.35 (14.10) | 19.42 (17.92) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 26.36 (17.76) | 29.95 (21.31) | 32.40 (19.24)
  Week 24 (n=24,15,28,15,43,55,51,0,40,20,24) | 35.21 (23.91) | 41.20 (19.27) | 22.50 (23.37) | 32.00 (19.13) | 30.26 (20.91) | 20.13 (16.50) | 19.06 (16.73) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 27.05 (17.55) | 24.05 (17.75) | 29.42 (21.01)

16. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PGA) of Arthritis Pain at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: as for outcome 15
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 50 | 17 | 46 | 59 | 57 | 53 | 44 | 57 | 25
mm
  Week 2 (n=54,0,50,0,46,59,57,53,0,57,0) | -9.83 (18.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -14.24 (19.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -14.93 (22.19) | -21.14 (20.74) | -22.21 (26.01) | -15.19 (19.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.00 (21.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,46,0,45,57,55,49,0,53,0) | -14.24 (18.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -21.93 (22.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -22.24 (21.63) | -26.61 (23.51) | -36.24 (26.36) | -18.65 (23.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.47 (25.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,47,0,44,58,55,48,0,52,0) | -22.10 (22.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -26.70 (23.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -26.36 (21.04) | -30.48 (22.57) | -38.24 (27.62) | -23.44 (21.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.38 (27.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,47,0,46,56,54,47,0,46,0) | -21.72 (21.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -25.53 (24.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -33.48 (22.13) | -31.88 (21.14) | -41.04 (26.88) | -24.45 (21.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -20.22 (25.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,48,0,45,56,53,45,0,46,0) | -20.04 (22.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -23.31 (24.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -32.20 (23.25) | -36.93 (23.90) | -42.70 (25.85) | -23.31 (24.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -19.41 (24.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,45,56,54,46,0,46,0) | -19.33 (20.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -24.57 (23.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -35.84 (20.73) | -36.50 (22.13) | -42.04 (24.60) | -25.74 (23.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -19.48 (27.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,29,17,45,55,53,0,43,20,25) | -28.11 (19.93) | -18.59 (24.63) | -31.24 (31.83) | -23.59 (17.14) | -35.60 (22.92) | -37.87 (21.09) | -44.66 (26.28) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -37.28 (19.72) | -35.15 (25.29) | -29.96 (23.75)
  Week 20 (n=27,16,28,16,44,51,53,0,44,19,25) | -25.44 (17.89) | -20.38 (20.91) | -33.29 (28.80) | -25.19 (18.46) | -38.55 (21.77) | -41.49 (18.87) | -47.11 (23.87) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -36.86 (20.07) | -32.89 (19.37) | -31.56 (24.08)
  Week 24 (n=24,15,27,15,42,54,51,0,40,20,24) | -24.38 (13.92) | -24.87 (25.37) | -34.78 (32.39) | -33.73 (17.12) | -35.55 (24.81) | -41.59 (18.94) | -47.12 (23.42) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -35.83 (22.06) | -39.80 (24.35) | -35.13 (23.70)

17. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 milligram per liter (mg/L) to 10 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 61 | 57 | 53 | 43 | 59 | 25
mg/L
  Baseline (n=54,0,51,0,49,61,57,53,0,59,0) | 21.39 (22.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.22 (19.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.51 (30.39) | 16.66 (16.85) | 21.70 (33.01) | 20.09 (23.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 23.53 (27.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=53,0,51,0,48,60,57,52,0,56,0) | 16.09 (17.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.63 (16.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.33 (17.71) | 4.37 (5.98) | 6.18 (9.45) | 9.54 (13.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.14 (36.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,48,0,45,57,53,49,0,53,0) | 16.81 (19.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.33 (13.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.32 (10.20) | 3.15 (5.93) | 5.04 (7.15) | 13.74 (19.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.69 (35.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=47,0,48,0,45,58,55,48,0,52,0) | 15.47 (16.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.76 (12.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.73 (9.80) | 4.00 (7.25) | 4.43 (6.21) | 15.47 (21.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.13 (33.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,56,53,47,0,45,0) | 21.80 (33.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.61 (26.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.22 (11.35) | 3.52 (5.82) | 4.50 (7.80) | 13.60 (18.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.06 (33.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,48,0,46,57,52,45,0,46,0) | 15.89 (21.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.20 (12.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.49 (10.77) | 2.34 (1.90) | 3.14 (4.45) | 14.31 (18.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.87 (36.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,45,54,52,45,0,45,0) | 16.89 (21.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.23 (12.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.13 (12.01) | 3.12 (3.48) | 3.62 (3.88) | 14.53 (20.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.00 (52.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,55,51,0,43,20,25) | 11.64 (15.98) | 9.86 (18.85) | 7.64 (11.06) | 9.21 (12.03) | 8.03 (16.57) | 4.65 (7.38) | 4.50 (7.05) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.73 (7.66) | 21.98 (28.43) | 6.04 (7.33)
  Week 20 (n=26,16,29,16,45,53,52,0,43,18,25) | 8.90 (7.91) | 4.02 (3.32) | 7.32 (8.75) | 7.20 (12.14) | 4.72 (4.57) | 2.85 (3.81) | 5.34 (9.65) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 6.82 (9.21) | 17.89 (15.34) | 4.65 (5.85)
  Week 24 (n=24,16,28,15,41,55,52,0,40,20,24) | 12.41 (13.51) | 10.51 (18.33) | 10.02 (15.12) | 5.74 (6.42) | 6.31 (7.79) | 5.65 (10.51) | 2.51 (2.50) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 6.01 (9.02) | 18.35 (17.49) | 5.39 (8.57)

18. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 mg/L to 10 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 53 | 17 | 51 | 17 | 48 | 60 | 57 | 52 | 43 | 56 | 25
mg/L
  Week 2 (n=53,0,51,0,48,60,57,52,0,56,0) | -5.59 (12.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.59 (11.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.32 (25.84) | -11.77 (16.87) | -15.53 (28.18) | -10.82 (17.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.63 (20.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,48,0,45,57,53,49,0,53,0) | -5.35 (15.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.84 (13.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.47 (27.76) | -13.88 (15.71) | -16.29 (32.42) | -6.73 (19.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.68 (30.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=47,0,48,0,45,58,55,48,0,52,0) | -7.04 (17.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.46 (15.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -18.20 (25.77) | -13.09 (18.13) | -17.78 (31.72) | -5.64 (21.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.13 (24.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,56,53,47,0,45,0) | -0.88 (34.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.61 (29.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.68 (26.27) | -12.70 (16.84) | -18.12 (33.97) | -7.65 (22.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.68 (25.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,48,0,46,57,52,45,0,46,0) | -7.41 (17.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.97 (16.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.80 (30.17) | -14.46 (17.28) | -19.68 (33.41) | -7.02 (21.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.60 (26.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,45,54,52,45,0,45,0) | -5.62 (19.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.79 (18.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.67 (27.63) | -13.28 (16.77) | -17.12 (29.92) | -7.29 (23.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.27 (45.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,55,51,0,43,20,25) | -5.08 (21.05) | -21.54 (34.58) | -4.63 (17.15) | -12.89 (23.41) | -15.57 (28.20) | -12.54 (19.07) | -18.41 (33.75) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -16.19 (25.25) | -0.54 (19.76) | -18.29 (27.14)
  Week 20 (n=26,16,29,16,45,53,52,0,43,18,25) | -8.39 (13.06) | -25.36 (28.34) | -5.33 (17.10) | -14.73 (25.04) | -19.21 (28.52) | -14.08 (17.85) | -17.67 (35.23) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -15.09 (25.59) | -6.87 (17.01) | -19.68 (30.10)
  Week 24 (n=24,16,28,15,41,55,52,0,40,20,24) | -4.19 (14.90) | -18.87 (31.77) | -2.25 (20.44) | -17.13 (26.10) | -19.43 (29.21) | -10.50 (19.53) | -20.43 (33.71) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -16.00 (25.94) | -4.18 (21.73) | -19.77 (30.92)

19. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 49 | 60 | 57 | 53 | 44 | 58 | 25
units on a scale
  Baseline (n=54,0,51,0,49,60,57,53,0,58,0) | 1.57 (0.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.53 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.40 (0.73) | 1.49 (0.74) | 1.62 (0.70) | 1.44 (0.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.54 (0.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,48,60,57,53,0,56,0) | 1.45 (0.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.28 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.22 (0.73) | 1.22 (0.68) | 1.26 (0.66) | 1.23 (0.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.49 (0.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,46,0,45,57,55,49,0,53,0) | 1.45 (0.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.23 (0.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.14 (0.67) | 1.04 (0.74) | 1.08 (0.68) | 1.31 (0.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.38 (0.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,44,59,54,48,0,52,0) | 1.30 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.24 (0.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.14 (0.71) | 1.00 (0.72) | 0.93 (0.71) | 1.19 (0.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.31 (0.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,46,57,54,47,0,46,0) | 1.29 (0.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.12 (0.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.99 (0.65) | 0.97 (0.75) | 0.86 (0.68) | 1.12 (0.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.24 (0.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,57,53,45,0,46,0) | 1.25 (0.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.20 (0.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.94 (0.75) | 0.86 (0.68) | 0.81 (0.71) | 1.18 (0.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.24 (0.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,57,54,46,0,46,0) | 1.28 (0.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.09 (0.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.94 (0.73) | 0.81 (0.68) | 0.78 (0.66) | 1.13 (0.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.24 (0.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,29,17,46,56,54,0,43,20,25) | 1.02 (0.72) | 1.34 (0.81) | 1.04 (0.79) | 1.31 (0.72) | 0.91 (0.74) | 0.85 (0.72) | 0.73 (0.63) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.95 (0.67) | 1.28 (0.66) | 0.86 (0.82)
  Week 20 (n=27,16,29,15,45,53,52,0,44,19,25) | 1.05 (0.71) | 1.20 (0.65) | 1.00 (0.78) | 1.04 (0.67) | 0.96 (0.76) | 0.80 (0.75) | 0.71 (0.65) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.95 (0.71) | 1.30 (0.69) | 0.82 (0.78)
  Week 24 (n=24,16,29,15,43,55,52,0,40,20,24) | 1.02 (0.65) | 1.29 (0.66) | 0.96 (0.83) | 1.00 (0.74) | 0.95 (0.81) | 0.81 (0.73) | 0.79 (0.67) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.93 (0.65) | 1.20 (0.81) | 0.69 (0.75)

20. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: as for outcome 19
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 59 | 57 | 53 | 44 | 56 | 24
units on a scale
  Week 2 (n=54,0,51,0,48,59,57,53,0,56,0) | -0.13 (0.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.25 (0.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.16 (0.47) | -0.27 (0.37) | -0.36 (0.63) | -0.21 (0.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.04 (0.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,46,0,45,56,55,49,0,52,0) | -0.14 (0.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.30 (0.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.26 (0.51) | -0.44 (0.60) | -0.55 (0.61) | -0.14 (0.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.09 (0.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=48,0,48,0,44,58,54,48,0,51,0) | -0.31 (0.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.28 (0.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.30 (0.56) | -0.49 (0.49) | -0.68 (0.73) | -0.25 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.17 (0.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,46,56,54,47,0,45,0) | -0.34 (0.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.40 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.37 (0.61) | -0.54 (0.60) | -0.73 (0.66) | -0.32 (0.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.24 (0.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,46,56,53,45,0,45,0) | -0.36 (0.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.34 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.45 (0.68) | -0.59 (0.56) | -0.78 (0.67) | -0.29 (0.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.24 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,56,54,46,0,45,0) | -0.30 (0.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.42 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.43 (0.65) | -0.63 (0.58) | -0.81 (0.71) | -0.32 (0.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.24 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,29,17,46,55,54,0,43,20,24) | -0.54 (0.63) | -0.29 (0.58) | -0.46 (0.55) | -0.31 (0.54) | -0.47 (0.66) | -0.60 (0.68) | -0.86 (0.67) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -0.49 (0.56) | -0.33 (0.52) | -0.55 (0.65)
  Week 20 (n=27,16,29,15,45,52,52,0,44,19,24) | -0.51 (0.73) | -0.35 (0.57) | -0.49 (0.56) | -0.51 (0.69) | -0.42 (0.66) | -0.62 (0.67) | -0.87 (0.68) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -0.50 (0.66) | -0.28 (0.39) | -0.59 (0.62)
  Week 24 (n=24,16,29,15,43,54,52,0,40,20,23) | -0.58 (0.67) | -0.26 (0.62) | -0.53 (0.59) | -0.56 (0.75) | -0.45 (0.75) | -0.63 (0.66) | -0.82 (0.67) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -0.53 (0.66) | -0.41 (0.60) | -0.72 (0.55)

21. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (<=) 3.2 implied low disease activity and greater than (>) 3.2 to 5.1 implied moderate to high disease activity, and less than (<) 2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adalimumab to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in adalimumab 40 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.Participants who administered Adalimumab initially were switched to CP-690,550 5 milligram (mg) tablet from Week 12 to Week 24.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 17 | 51 | 17 | 48 | 59 | 57 | 52 | 43 | 58 | 25
units on a scale
  Baseline (n=54,0,51,0,47,59,57,52,0,58,0) | 5.51 (0.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.37 (0.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.58 (0.88) | 5.46 (0.82) | 5.46 (0.96) | 5.35 (0.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.62 (0.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=53,0,51,0,48,60,57,52,0,56,0) | 4.96 (1.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.60 (1.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.63 (1.15) | 4.16 (0.96) | 4.32 (1.09) | 4.59 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.24 (1.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,45,57,53,49,0,53,0) | 4.77 (1.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.16 (1.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.36 (1.00) | 3.71 (1.15) | 3.71 (1.09) | 4.40 (1.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.01 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=47,0,48,0,45,58,55,48,0,52,0) | 4.42 (1.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.02 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.16 (1.06) | 3.45 (1.11) | 3.34 (1.29) | 4.19 (1.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.92 (1.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,56,53,47,0,45,0) | 4.52 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.00 (1.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.01 (1.25) | 3.37 (1.06) | 3.13 (1.21) | 4.23 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.84 (1.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,48,0,46,57,52,45,0,46,0) | 4.37 (1.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.92 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.80 (1.21) | 3.06 (0.98) | 3.05 (1.18) | 4.12 (1.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.83 (1.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,45,54,52,45,0,45,0) | 4.57 (1.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.96 (1.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.76 (1.38) | 3.11 (1.18) | 3.06 (1.13) | 4.13 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.83 (1.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,55,51,0,43,20,25) | 3.63 (1.35) | 4.47 (1.13) | 3.30 (1.07) | 4.75 (1.16) | 3.55 (1.41) | 3.06 (1.13) | 2.92 (1.14) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 3.32 (1.13) | 3.93 (1.22) | 4.01 (1.08)
  Week 20 (n=26,16,29,16,45,53,52,0,43,18,25) | 3.94 (1.40) | 4.14 (0.92) | 3.26 (1.00) | 4.44 (1.32) | 3.68 (1.38) | 2.85 (1.10) | 2.93 (1.20) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 3.33 (1.17) | 3.97 (1.08) | 3.78 (1.11)
  Week 24 (n=24,16,28,15,41,55,52,0,39,20,24) | 4.11 (1.26) | 4.42 (1.12) | 3.11 (1.25) | 4.33 (1.28) | 3.64 (1.22) | 2.92 (1.03) | 2.82 (1.17) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 3.40 (1.17) | 3.96 (1.36) | 3.61 (1.13)

22. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Week 2, 4, 6, 8, 10, 12, 16, 20 and 24/ET
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and > 3.2 to 5.1 implied moderate to high disease activity, and < 2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 53 | 17 | 51 | 17 | 46 | 58 | 57 | 51 | 43 | 55 | 24
units on a scale
  Week 2 (n=53,0,51,0,46,58,57,51,0,55,0) | -0.55 (0.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.77 (0.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.95 (0.85) | -1.28 (0.99) | -1.14 (1.03) | -0.73 (0.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.37 (0.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,47,0,43,56,53,48,0,52,0) | -0.75 (1.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.17 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.26 (0.95) | -1.75 (1.23) | -1.72 (1.27) | -0.91 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.63 (0.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=47,0,48,0,43,56,55,47,0,51,0) | -1.17 (1.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.31 (1.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.50 (0.95) | -1.99 (1.25) | -2.14 (1.44) | -1.12 (1.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.73 (1.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,45,54,53,46,0,44,0) | -1.09 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.34 (1.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.60 (1.09) | -2.05 (1.13) | -2.31 (1.44) | -1.08 (1.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.84 (1.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,48,0,44,56,52,44,0,45,0) | -1.24 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.43 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.87 (1.18) | -2.40 (1.12) | -2.41 (1.25) | -1.23 (1.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.76 (1.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,43,53,52,44,0,44,0) | -1.04 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.36 (1.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.87 (1.29) | -2.29 (1.25) | -2.37 (1.26) | -1.18 (1.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.80 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,44,54,51,0,43,20,24) | -1.83 (1.25) | -1.36 (1.07) | -1.80 (1.19) | -0.95 (0.96) | -2.05 (1.33) | -2.41 (1.20) | -2.49 (1.31) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -2.01 (1.12) | -1.73 (1.19) | -1.54 (1.16)
  Week 20 (n=26,16,29,16,43,52,52,0,43,18,24) | -1.52 (1.39) | -1.61 (1.23) | -1.96 (1.18) | -1.25 (1.13) | -1.96 (1.33) | -2.54 (1.17) | -2.52 (1.40) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -2.01 (1.07) | -1.77 (0.91) | -1.76 (1.27)
  Week 24 (n=24,16,28,15,39,54,52,0,39,20,23) | -1.27 (1.22) | -1.33 (1.36) | -2.08 (1.34) | -1.28 (1.02) | -2.07 (1.24) | -2.51 (1.20) | -2.62 (1.47) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -1.94 (1.29) | -1.71 (1.26) | -2.04 (1.43)

23. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and PtGA of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implies low disease activity and > 3.2 to 5.1 implies moderate to high disease activity, and < 2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 51 | 17 | 50 | 17 | 47 | 60 | 54 | 51 | 43 | 56 | 24
units on a scale
  Baseline (n=49,0,49,0,47,59,54,51,0,56,0) | 6.51 (0.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.35 (0.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.57 (0.87) | 6.46 (0.85) | 6.46 (0.95) | 6.30 (0.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.56 (0.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=51,0,50,0,47,60,54,51,0,53,0) | 5.92 (1.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.57 (1.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.61 (1.34) | 5.20 (1.07) | 5.20 (1.29) | 5.53 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.04 (1.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=49,0,46,0,46,57,53,46,0,51,0) | 5.73 (1.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.10 (1.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.23 (1.09) | 4.69 (1.31) | 4.46 (1.43) | 5.22 (1.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.70 (1.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=46,0,47,0,45,58,54,47,0,51,0) | 5.36 (1.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.91 (1.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.90 (1.19) | 4.33 (1.32) | 4.02 (1.57) | 4.99 (1.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.64 (1.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,48,0,47,56,54,46,0,44,0) | 5.31 (1.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.89 (1.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.70 (1.24) | 4.22 (1.18) | 3.80 (1.45) | 5.01 (1.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.56 (1.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,49,0,45,56,53,43,0,44,0) | 5.22 (1.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.81 (1.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.50 (1.31) | 3.93 (1.17) | 3.71 (1.31) | 4.98 (1.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.54 (1.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,46,56,53,45,0,45,0) | 5.41 (1.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.78 (1.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.37 (1.43) | 3.95 (1.38) | 3.77 (1.32) | 5.00 (1.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.39 (1.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,45,55,54,0,42,20,24) | 4.39 (1.33) | 5.36 (1.23) | 3.96 (1.31) | 5.70 (1.22) | 4.25 (1.47) | 3.86 (1.36) | 3.63 (1.39) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 4.08 (1.19) | 4.53 (1.34) | 4.95 (1.30)
  Week 20 (n=26,16,29,16,45,51,52,0,43,19,24) | 4.76 (1.50) | 5.22 (0.93) | 4.08 (1.30) | 5.31 (1.37) | 4.47 (1.47) | 3.67 (1.39) | 3.54 (1.29) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 4.04 (1.35) | 4.47 (1.50) | 4.62 (1.27)
  Week 24 (n=24,16,29,15,43,54,51,0,38,20,23) | 4.87 (1.43) | 5.27 (1.42) | 3.72 (1.58) | 5.19 (1.23) | 4.33 (1.40) | 3.62 (1.26) | 3.61 (1.31) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 4.22 (1.26) | 4.51 (1.41) | 4.28 (1.20)

24. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR [mm/hour] and PtGA of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implies low disease activity and > 3.2 to 5.1 implies moderate to high disease activity, and < 2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 48 | 15 | 49 | 16 | 45 | 58 | 52 | 50 | 42 | 53 | 22
units on a scale
  Week 2 (n=48,0,49,0,45,58,52,50,0,53,0) | -0.56 (1.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.81 (1.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.98 (0.88) | -1.32 (1.05) | -1.27 (1.28) | -0.82 (1.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.53 (1.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=46,0,45,0,44,55,51,45,0,50,0) | -0.82 (1.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.29 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.31 (0.89) | -1.81 (1.32) | -1.95 (1.50) | -1.14 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.87 (1.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=43,0,46,0,43,56,52,46,0,49,0) | -1.26 (1.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.41 (1.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.67 (0.97) | -2.16 (1.40) | -2.39 (1.58) | -1.29 (1.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.97 (1.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=43,0,46,0,45,54,52,45,0,42,0) | -1.30 (1.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.40 (1.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.84 (0.99) | -2.28 (1.21) | -2.63 (1.56) | -1.29 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.00 (1.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=42,0,47,0,43,54,51,42,0,42,0) | -1.37 (1.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.48 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.05 (1.28) | -2.55 (1.30) | -2.78 (1.42) | -1.37 (1.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.00 (1.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=40,0,44,0,44,54,51,44,0,43,0) | -1.16 (1.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.52 (1.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.16 (1.32) | -2.55 (1.46) | -2.65 (1.41) | -1.35 (1.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.17 (1.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=25,15,29,16,43,53,52,0,41,20,22) | -1.97 (1.42) | -1.51 (1.08) | -2.06 (1.38) | -1.18 (0.93) | -2.30 (1.29) | -2.63 (1.37) | -2.83 (1.53) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -2.29 (1.15) | -1.97 (1.28) | -1.63 (0.93)
  Week 20 (n=24,15,28,15,43,49,50,0,42,19,22) | -1.54 (1.58) | -1.58 (1.34) | -2.02 (1.37) | -1.47 (1.15) | -2.02 (1.34) | -2.68 (1.29) | -2.88 (1.46) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -2.33 (1.28) | -2.03 (1.11) | -1.91 (1.03)
  Week 24 (n=22,15,28,14,41,52,49,0,37,20,21) | -1.33 (1.46) | -1.58 (1.58) | -2.38 (1.50) | -1.51 (1.04) | -2.24 (1.31) | -2.79 (1.37) | -2.78 (1.52) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -2.08 (1.32) | -1.99 (1.27) | -2.30 (1.24)

25. Secondary Outcome: Percentage of Participants With Disease Improvement Based on DAS28-4 (ESR)
Description: Disease improvement was classified as good, moderate, and none based on improvement in DAS28-4 (ESR) from baseline and present DAS28-4 (ESR) score. Good: an improvement from baseline of >1.2 and a present score of <=3.2; none: an improvement of <=0.6 or >0.6 to <=1.2 with a present score of >5.1; remaining participants were classified as having moderate (Mod) improvement. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ET
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 51 | 17 | 50 | 17 | 47 | 60 | 54 | 51 | 43 | 53 | 24
percentage of participants
  Week 2: Good (n=51,0,50,0,47,60,54,51,0,53,0) | 3.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.3 | 3.3 | 7.4 | 3.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Mod (n=51,0,50,0,47,60,54,51,0,53,0) | 13.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.9 | 53.3 | 42.6 | 39.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: None (n=51,0,50,0,47,60,54,51,0,53,0) | 76.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 68.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 59.6 | 40.0 | 46.3 | 54.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 73.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: Good (n=49,0,46,0,46,57,53,46,0,51,0) | 2.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.2 | 14.0 | 17.0 | 10.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: Mod (n=49,0,46,0,46,57,53,46,0,51,0) | 28.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 56.5 | 52.6 | 50.9 | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: None (n=49,0,46,0,46,57,53,46,0,51,0) | 63.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.0 | 29.8 | 28.3 | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: Good (n=46,0,47,0,45,58,54,47,0,51,0) | 2.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.2 | 22.4 | 29.6 | 14.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: Mod (n=46,0,47,0,45,58,54,47,0,51,0) | 47.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 66.7 | 53.4 | 50.0 | 42.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: None (n=46,0,47,0,45,58,54,47,0,51,0) | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.7 | 20.7 | 16.7 | 40.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: Good (n=47,0,48,0,47,56,54,46,0,44,0) | 6.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.5 | 17.9 | 37.0 | 10.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: Mod (n=47,0,48,0,47,56,54,46,0,44,0) | 44.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 68.1 | 64.3 | 40.7 | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: None (n=47,0,48,0,47,56,54,46,0,44,0) | 40.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 19.1 | 14.3 | 18.5 | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 52.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10: Good (n=46,0,49,0,45,56,53,43,0,44,0) | 8.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.6 | 25.0 | 41.5 | 9.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10: Mod (n=46,0,49,0,45,56,53,43,0,44,0) | 45.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 55.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 57.8 | 60.7 | 45.3 | 46.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10: None (n=46,0,49,0,45,56,53,43,0,44,0) | 37.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.2 | 10.7 | 9.4 | 41.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Good (n=44,0,46,0,46,56,53,45,0,45,0) | 9.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.7 | 32.1 | 37.7 | 11.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mod (n=44,0,46,0,46,56,53,45,0,45,0) | 31.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.3 | 50.0 | 47.2 | 42.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: None (n=44,0,46,0,46,56,53,45,0,45,0) | 50.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 19.6 | 14.3 | 11.3 | 44.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16: Good (n=27,17,30,17,45,55,54,0,42,20,24) | 18.5 | 5.9 | 26.7 | 5.9 | 22.2 | 32.7 | 44.4 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 23.8 | 20.0 | 8.3
  Week 16: Mod (n=27,17,30,17,45,55,54,0,42,20,24) | 44.4 | 52.9 | 50.0 | 35.3 | 60.0 | 52.7 | 40.7 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 61.9 | 50.0 | 54.2
  Week 16: None (n=27,17,30,17,45,55,54,0,42,20,24) | 29.6 | 29.4 | 20.0 | 52.9 | 13.3 | 10.9 | 11.1 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 11.9 | 30.0 | 29.2
  Week 20: Good (n=26,16,29,16,45,51,52,0,43,19,24) | 11.5 | 0.0 | 27.6 | 0.0 | 20.0 | 37.3 | 38.5 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 27.9 | 26.3 | 12.5
  Week 20: Mod (n=26,16,29,16,45,51,52,0,43,19,24) | 42.3 | 56.3 | 55.2 | 62.5 | 48.9 | 52.9 | 48.1 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 60.5 | 47.4 | 62.5
  Week 20: None (n=26,16,29,16,45,51,52,0,43,19,24) | 38.5 | 37.5 | 13.8 | 31.3 | 26.7 | 5.9 | 9.6 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 9.3 | 26.3 | 16.7
  Week 24: Good (n=24,16,29,15,43,54,51,0,38,20,23) | 12.5 | 12.5 | 41.4 | 6.7 | 20.9 | 38.9 | 43.1 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 23.7 | 20.0 | 8.7
  Week 24: Mod (n=24,16,29,15,43,54,51,0,38,20,23) | 37.5 | 43.8 | 41.4 | 60.0 | 58.1 | 48.1 | 45.1 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 57.9 | 60.0 | 65.2
  Week 24: None (n=24,16,29,15,43,54,51,0,38,20,23) | 41.7 | 37.5 | 13.8 | 26.7 | 16.3 | 9.3 | 7.8 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 15.8 | 20.0 | 17.4

26. Secondary Outcome: Percentage of Participants With Disease Remission Based on Normal C-reactive Protein (CRP)
Description: CRP value less than or equal to upper limit of normal (ULN) implied disease remission (ULN=4.9 mg/L).
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ ET
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 43 | 17 | 33 | 17 | 40 | 45 | 39 | 40 | 43 | 37 | 25
percentage of participants
  Week 2 (n=43,0,33,0,40,45,39,40,0,37,0) | 25.58 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 62.50 | 71.11 | 66.67 | 40.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.70 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=40,0,30,0,37,43,37,37,0,35,0) | 30.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 62.16 | 83.72 | 62.16 | 35.14 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.71 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=39,0,30,0,39,44,37,36,0,34,0) | 20.51 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 56.41 | 79.55 | 67.57 | 30.56 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.88 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=39,0,30,0,39,42,36,35,0,31,0) | 25.64 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 66.67 | 78.57 | 75.00 | 25.71 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.68 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=38,0,30,0,38,43,34,33,0,30,0) | 26.32 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 53.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 65.79 | 90.70 | 79.41 | 21.21 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=36,0,28,0,37,41,35,33,0,30,0) | 22.22 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.86 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 62.16 | 75.61 | 68.57 | 30.30 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,55,51,0,43,20,25) | 48.1 | 41.2 | 53.3 | 64.7 | 69.6 | 78.2 | 82.4 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 67.4 | 35.0 | 68.0
  Week 20 (n=26,16,29,16,45,53,52,0,43,18,25) | 46.2 | 75.0 | 58.6 | 75.0 | 68.9 | 88.7 | 76.9 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 67.4 | 16.7 | 72.0
  Week 24 (n=24,16,28,15,41,55,52,0,40,20,24) | 33.3 | 75.0 | 46.4 | 60.0 | 65.9 | 72.7 | 84.6 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 72.5 | 30.0 | 66.7

27. Secondary Outcome: Percentage of Participants With Disease Remission Based on DAS28-3 (CRP)
Description: DAS28-3 (CRP) defined remission was classified as a score of <2.6.
Time Frame: Week 2, 4, 6, 8, 10, 12, 16, 20, 24/ ET
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 53 | 17 | 50 | 17 | 48 | 60 | 57 | 52 | 43 | 56 | 25
percentage of participants
  Week 2 (n=53,0,50,0,48,60,57,52,0,56,0) | 1.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.17 | 5.00 | 7.02 | 1.92 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=50,0,46,0,45,57,53,49,0,53,0) | 6.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.52 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.44 | 17.54 | 15.09 | 12.24 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=47,0,47,0,45,58,55,48,0,52,0) | 8.51 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.77 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.89 | 24.14 | 32.73 | 12.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.92 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=47,0,47,0,47,56,53,47,0,45,0) | 2.13 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.77 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.89 | 21.43 | 41.51 | 12.77 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.44 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 10 (n=46,0,47,0,46,57,52,45,0,46,0) | 10.87 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.51 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.74 | 31.58 | 38.46 | 15.56 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.35 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,45,0,45,54,52,45,0,45,0) | 9.30 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.89 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.44 | 33.33 | 40.38 | 4.44 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=27,17,30,17,46,55,51,0,43,20,25) | 22.2 | 5.9 | 30.0 | 5.9 | 28.3 | 36.4 | 43.1 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 25.6 | 15.0 | 12.0
  Week 20 (n=26,16,29,16,45,53,52,0,43,18,25) | 19.2 | 6.3 | 20.7 | 6.3 | 20.0 | 43.4 | 42.3 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 25.6 | 5.6 | 12.0
  Week 24 (n=24,16,28,15,41,55,52,0,39,20,24) | 16.7 | 6.3 | 39.3 | 6.7 | 22.0 | 36.4 | 50.0 | NA — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 23.1 | 15.0 | 25.0

28. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 domains (of 2 components [C]; physical [Ph] and mental [Mn]) of functional health and well being: physical and social (So) functioning (Fn), physical and emotional role (role-physical [R-P], role-emotional [R-E]) limitations, bodily pain (BP), general health (GH), vitality (Vit), mental health (MnH). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 15 | 51 | 15 | 49 | 61 | 57 | 53 | 40 | 59 | 24
units on a scale
  Baseline: Ph Fn (n=54,0,51,0,49,61,57,53,0,59,0) | 29.75 (10.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.88 (11.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.93 (11.75) | 30.30 (10.65) | 30.08 (9.66) | 30.55 (8.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.25 (9.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: R-P (n=54,0,51,0,49,61,57,53,0,59,0) | 32.82 (9.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.21 (9.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.31 (10.46) | 31.44 (9.32) | 31.63 (8.07) | 32.87 (10.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.20 (8.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: BP (n=54,0,51,0,49,61,57,53,0,59,0) | 32.60 (7.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.41 (8.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.21 (7.30) | 33.48 (6.48) | 32.54 (7.25) | 32.23 (6.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.19 (8.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: GH (n=54,0,51,0,49,61,56,53,0,59,0) | 34.80 (8.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.60 (8.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.89 (8.57) | 34.24 (8.23) | 34.58 (8.81) | 35.55 (9.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.35 (7.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Vit (n=54,0,51,0,49,61,57,53,0,59,0) | 40.30 (10.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.46 (11.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.28 (10.95) | 38.94 (10.43) | 38.34 (10.70) | 36.42 (10.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.87 (9.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: So Fn (n=54,0,51,0,49,61,57,53,0,59,0) | 36.35 (11.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.17 (11.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.14 (10.88) | 35.93 (10.73) | 36.28 (12.11) | 33.28 (10.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.50 (10.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: R-E (n=54,0,51,0,49,61,57,53,0,59,0) | 33.28 (11.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.09 (12.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.14 (11.74) | 34.40 (14.35) | 32.21 (12.92) | 32.26 (12.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.21 (14.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: MnH (n=54,0,51,0,49,61,57,53,0,59,0) | 39.16 (11.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.58 (11.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.94 (12.02) | 37.73 (12.10) | 37.80 (12.62) | 36.22 (12.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.45 (11.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Ph C (n=54,0,51,0,49,61,56,53,0,59,0) | 31.49 (7.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.52 (9.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.12 (9.52) | 31.44 (8.16) | 31.82 (7.59) | 32.67 (7.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.94 (6.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Mn C (n=54,0,51,0,49,61,56,53,0,59,0) | 40.23 (11.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.47 (11.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.52 (11.82) | 39.56 (12.17) | 38.64 (12.45) | 36.46 (12.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.96 (12.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph Fn (n=44,0,46,0,45,57,54,45,0,46,0) | 32.59 (11.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.48 (11.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.36 (10.74) | 39.42 (11.99) | 38.44 (11.65) | 35.61 (10.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.11 (11.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-P (n=44,0,46,0,45,57,54,45,0,46,0) | 37.60 (8.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.27 (10.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.00 (9.31) | 40.78 (10.67) | 41.75 (11.45) | 36.83 (10.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.21 (9.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: BP (n=44,0,46,0,45,57,54,45,0,46,0) | 39.14 (7.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.87 (9.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.26 (9.13) | 45.65 (9.40) | 46.24 (10.30) | 37.67 (9.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.50 (9.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: GH (n=44,0,46,0,45,57,54,45,0,46,0) | 38.99 (7.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.45 (9.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.00 (7.90) | 40.11 (11.10) | 40.80 (11.07) | 38.42 (11.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.05 (8.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Vit (n=44,0,46,0,45,57,54,45,0,46,0) | 45.92 (10.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.37 (10.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.22 (10.15) | 48.59 (11.74) | 49.20 (11.73) | 44.88 (10.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.20 (11.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: So Fn (n=44,0,46,0,45,57,54,45,0,46,0) | 41.11 (11.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.55 (11.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.15 (9.20) | 43.93 (11.78) | 44.43 (12.15) | 38.43 (12.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.44 (11.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-E (n=44,0,46,0,45,57,53,45,0,46,0) | 37.86 (10.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.03 (13.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.98 (10.35) | 39.72 (12.80) | 39.23 (13.39) | 39.98 (12.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.23 (12.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: MnH (n=44,0,46,0,45,57,54,45,0,46,0) | 43.61 (11.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.50 (11.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.44 (10.86) | 43.29 (12.68) | 43.91 (13.60) | 42.94 (12.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.89 (10.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph C (n=44,0,46,0,45,57,53,45,0,46,0) | 35.76 (7.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.17 (8.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.15 (9.30) | 41.89 (9.70) | 42.44 (9.71) | 35.89 (10.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.00 (9.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mn C (n=44,0,46,0,45,57,53,45,0,46,0) | 45.03 (11.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.82 (11.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.49 (9.96) | 44.46 (12.89) | 44.91 (14.05) | 44.22 (12.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.22 (10.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: Ph Fn (n=24,15,29,15,43,55,52,0,40,20,24) | 35.64 (10.40) | 35.57 (11.72) | 37.66 (12.25) | 33.32 (12.79) | 36.23 (12.04) | 40.43 (11.67) | 39.67 (10.91) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 38.36 (10.74) | 34.94 (10.76) | 41.60 (10.62)
  Week 24: R-P (n=24,15,29,15,43,55,52,0,40,20,24) | 37.06 (9.13) | 39.38 (10.26) | 42.33 (9.00) | 34.98 (9.64) | 39.82 (11.02) | 41.80 (10.75) | 41.17 (9.61) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 38.98 (9.51) | 37.14 (9.88) | 43.38 (9.50)
  Week 24: BP (n=24,15,29,15,43,55,52,0,40,20,24) | 39.26 (8.99) | 38.11 (9.41) | 42.15 (10.95) | 41.89 (9.03) | 42.05 (10.07) | 46.73 (10.09) | 45.37 (9.66) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 42.66 (9.22) | 39.91 (7.67) | 43.96 (10.01)
  Week 24: GH (n=24,15,29,15,43,55,52,0,40,20,24) | 41.20 (10.49) | 38.47 (8.43) | 42.53 (10.23) | 37.11 (7.14) | 39.56 (8.79) | 41.46 (11.85) | 39.63 (10.19) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 39.62 (9.20) | 38.16 (8.74) | 42.84 (9.18)
  Week 24: Vit (n=24,15,29,15,43,55,52,0,40,20,24) | 45.85 (12.21) | 44.18 (8.74) | 49.29 (9.71) | 45.78 (9.47) | 46.28 (10.00) | 47.61 (11.24) | 46.51 (10.98) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 46.24 (9.33) | 46.47 (10.70) | 49.10 (9.72)
  Week 24: So Fn (n=24,15,29,15,43,55,52,0,40,20,24) | 42.08 (11.31) | 39.40 (9.26) | 44.25 (9.46) | 40.12 (8.86) | 41.76 (10.16) | 44.26 (12.32) | 42.69 (11.39) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 41.71 (9.99) | 41.85 (8.28) | 47.08 (9.37)
  Week 24: R-E (n=24,15,29,15,43,55,52,0,40,20,24) | 36.12 (13.51) | 39.03 (13.44) | 43.14 (10.38) | 32.81 (13.42) | 38.97 (12.29) | 40.82 (12.85) | 40.33 (11.52) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 41.20 (11.66) | 38.39 (10.81) | 42.27 (10.38)
  Week 24: MnH (n=24,15,29,15,43,55,52,0,40,20,24) | 45.55 (10.60) | 41.00 (8.92) | 44.76 (11.28) | 39.87 (8.37) | 43.20 (11.53) | 44.63 (12.75) | 43.08 (13.13) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 44.94 (10.13) | 43.53 (11.34) | 45.55 (11.08)
  Week 24: Ph C (n=24,15,29,15,43,55,52,0,40,20,24) | 37.35 (8.62) | 37.51 (9.25) | 40.21 (10.21) | 37.35 (9.07) | 39.03 (9.96) | 42.81 (9.89) | 41.80 (10.03) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 39.03 (9.50) | 36.55 (9.64) | 42.87 (9.13)
  Week 24: Mn C (n=24,15,29,15,43,55,52,0,40,20,24) | 44.79 (12.57) | 42.61 (9.01) | 47.43 (9.51) | 40.65 (8.04) | 44.18 (10.91) | 44.97 (12.87) | 43.73 (12.76) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 45.53 (10.29) | 45.01 (10.13) | 46.93 (10.63)

29. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Week 12 and 24/ET
Description: as for outcome 28
Time Frame: Baseline, Week 12, 24/ ET
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 44 | 15 | 46 | 15 | 45 | 57 | 54 | 45 | 40 | 46 | 24
units on a scale
  Week 12: Ph Fn (n=44,0,46,0,45,57,54,45,0,46,0) | 3.11 (11.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.90 (8.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.64 (10.60) | 8.90 (9.85) | 8.18 (10.11) | 5.05 (8.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.83 (9.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-P (n=44,0,46,0,45,57,54,45,0,46,0) | 4.34 (10.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.01 (9.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.64 (9.87) | 8.98 (9.94) | 9.71 (11.64) | 3.43 (12.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.84 (9.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: BP (n=44,0,46,0,45,57,54,45,0,46,0) | 6.36 (8.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.37 (9.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.15 (8.40) | 12.06 (9.21) | 13.73 (10.95) | 5.91 (8.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.91 (8.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: GH (n=44,0,46,0,45,57,53,45,0,46,0) | 3.46 (7.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.59 (8.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.21 (7.48) | 6.00 (8.92) | 6.63 (9.64) | 4.05 (9.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.41 (6.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Vit (n=44,0,46,0,45,57,54,45,0,46,0) | 5.25 (9.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.87 (9.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.76 (8.93) | 9.75 (11.53) | 10.75 (12.76) | 8.12 (10.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.73 (10.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: So Fn (n=44,0,46,0,45,57,54,45,0,46,0) | 12.71 (1.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.31 (1.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.03 (1.50) | 11.91 (1.58) | 13.88 (1.89) | 14.01 (2.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.71 (1.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-E (n=44,0,46,0,45,57,53,45,0,46,0) | 5.12 (12.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.70 (12.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.53 (13.45) | 5.86 (11.48) | 5.94 (14.19) | 6.82 (15.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.17 (13.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: MnH (n=44,0,46,0,45,57,54,45,0,46,0) | 4.86 (11.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.12 (9.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.13 (11.63) | 6.08 (8.39) | 5.42 (14.02) | 7.48 (10.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.00 (10.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph C (n=44,0,46,0,45,57,52,45,0,46,0) | 3.78 (7.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.96 (8.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.29 (7.95) | 10.01 (9.31) | 10.70 (9.83) | 3.47 (8.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.43 (9.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mn C (n=44,0,46,0,45,57,52,45,0,46,0) | 5.23 (10.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.33 (9.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.45 (11.77) | 5.38 (9.61) | 6.12 (13.57) | 7.59 (11.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.74 (9.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: Ph Fn (n=24,15,29,15,43,55,52,0,40,20,24) | 5.52 (8.28) | 7.30 (10.84) | 5.01 (10.60) | 6.87 (9.85) | 6.12 (11.54) | 9.60 (9.63) | 9.67 (11.58) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 7.21 (9.80) | 6.63 (7.01) | 7.80 (11.06)
  Week 24: R-P (n=24,15,29,15,43,55,52,0,40,20,24) | 4.39 (12.06) | 6.86 (9.49) | 7.18 (9.00) | 3.65 (11.91) | 7.18 (9.19) | 10.02 (11.19) | 9.37 (9.78) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.14 (12.41) | 6.61 (7.95) | 8.98 (9.30)
  Week 24: BP (n=24,15,29,15,43,55,52,0,40,20,24) | 4.65 (10.48) | 7.86 (11.86) | 7.40 (9.78) | 8.93 (9.70) | 9.89 (9.07) | 13.19 (9.64) | 13.13 (10.51) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 10.51 (9.55) | 6.23 (7.24) | 11.11 (10.03)
  Week 24: GH (n=24,15,29,15,43,55,51,0,40,20,24) | 4.23 (11.06) | 5.91 (8.60) | 5.10 (8.04) | 2.51 (7.65) | 5.64 (7.18) | 7.37 (9.15) | 5.44 (9.03) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.77 (8.35) | 5.46 (6.54) | 6.87 (10.73)
  Week 24: Vit (n=24,15,29,15,43,55,52,0,40,20,24) | 3.38 (9.20) | 8.12 (10.00) | 5.49 (9.01) | 8.46 (12.53) | 6.75 (8.31) | 9.20 (10.89) | 8.17 (12.01) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 9.13 (10.13) | 7.80 (10.10) | 9.37 (7.92)
  Week 24: So Fn (n=24,15,29,15,43,55,52,0,40,20,24) | 4.54 (11.10) | 7.27 (12.82) | 2.07 (11.61) | 7.64 (7.38) | 6.21 (11.51) | 7.93 (12.46) | 6.61 (13.46) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 7.77 (13.47) | 10.36 (10.15) | 10.23 (9.69)
  Week 24: R-E (n=24,15,29,15,43,55,52,0,40,20,24) | 2.75 (16.15) | 7.77 (14.09) | 6.43 (9.13) | 3.11 (13.72) | 4.70 (10.37) | 7.07 (14.41) | 7.55 (11.09) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 7.77 (16.06) | 6.22 (16.32) | 7.45 (12.18)
  Week 24: MnH (n=24,15,29,15,43,55,52,0,40,20,24) | 5.28 (8.92) | 7.51 (10.73) | 3.50 (9.18) | 5.44 (7.33) | 5.37 (13.10) | 7.68 (8.32) | 4.55 (13.22) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 9.19 (12.03) | 5.63 (10.81) | 7.86 (10.14)
  Week 24: Ph C (n=24,15,29,15,43,55,51,0,40,20,24) | 4.78 (7.89) | 6.50 (7.44) | 6.40 (9.31) | 6.05 (10.51) | 7.72 (9.12) | 10.77 (9.80) | 10.58 (10.83) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 6.32 (9.21) | 6.18 (6.21) | 8.73 (9.45)
  Week 24: Mn C (n=24,15,29,15,43,55,51,0,40,20,24) | 3.45 (9.84) | 7.51 (11.20) | 3.50 (7.24) | 5.10 (8.70) | 4.57 (11.28) | 6.25 (10.22) | 4.23 (12.36) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 8.67 (12.28) | 7.03 (12.02) | 7.91 (10.04)

30. Secondary Outcome: Euro Quality of Life 5 Dimension (EQ-5D)-Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 15 | 51 | 14 | 49 | 61 | 57 | 53 | 40 | 59 | 24
units on a scale
  Baseline (n=54,0,51,0,49,61,57,53,0,59,0) | 0.41 (0.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.33 (0.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.39 (0.37) | 0.41 (0.30) | 0.34 (0.35) | 0.36 (0.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.38 (0.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=43,0,46,0,45,56,54,45,0,45,0) | 0.56 (0.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.50 (0.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.60 (0.27) | 0.68 (0.25) | 0.66 (0.27) | 0.51 (0.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.53 (0.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=24,15,29,14,43,55,52,0,40,20,24) | 0.64 (0.23) | 0.55 (0.30) | 0.67 (0.22) | 0.58 (0.25) | 0.61 (0.30) | 0.68 (0.26) | 0.67 (0.26) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.60 (0.24) | 0.63 (0.22) | 0.73 (0.17)

31. Secondary Outcome: Change From Baseline in Euro Quality of Life 5 Dimension (EQ-5D)- Health State Profile Utility Score at Week 12 and 24/ET
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 43 | 15 | 46 | 14 | 45 | 56 | 54 | 45 | 40 | 45 | 24
units on a scale
  Week 12 (n=43,0,46,0,45,56,54,45,0,45,0) | 0.15 (0.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.14 (0.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.21 (0.33) | 0.27 (0.29) | 0.30 (0.37) | 0.16 (0.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.11 (0.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=24,15,29,14,43,55,52,0,40,20,24) | 0.23 (0.33) | 0.15 (0.34) | 0.23 (0.28) | 0.36 (0.36) | 0.23 (0.32) | 0.27 (0.31) | 0.32 (0.40) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.24 (0.36) | 0.21 (0.28) | 0.32 (0.28)

32. Other Pre Specified Outcome: Serum Immunoglobulin G (IgG), Immunoglobulin M (IgM) and Immunoglobulin A (IgA) Levels
Description: Blood samples for immunoglobulin assessments were obtained to determine IgG, IgM, and IgA levels in serum.
Time Frame: Baseline, Week 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 50 | 15 | 47 | 12 | 45 | 58 | 53 | 49 | 34 | 54 | 22
milligram per deciliter (mg/dL)
  Baseline: IgG (n=50,0,47,0,45,58,53,49,0,54,0) | 1261.68 (331.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1157.79 (290.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1219.31 (326.92) | 1219.38 (397.93) | 1157.57 (271.58) | 1143.78 (359.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1221.28 (402.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: IgM (n=50,0,47,0,45,58,53,49,0,54,0) | 154.20 (77.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 172.81 (72.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 115.04 (48.12) | 160.69 (75.04) | 156.04 (73.34) | 144.27 (103.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 169.78 (83.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: IgA (n=50,0,47,0,45,58,51,49,0,54,0) | 356.76 (242.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 285.34 (121.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 321.58 (171.12) | 316.60 (140.26) | 304.14 (164.97) | 323.49 (134.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 327.00 (177.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: IgG (n=21,15,24,12,35,48,44,0,34,17,22) | 1207.57 (330.54) | 1148.07 (439.24) | 1068.08 (266.71) | 1142.75 (315.33) | 1169.97 (280.16) | 1111.42 (286.08) | 1073.66 (274.31) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 1143.91 (290.22) | 1153.76 (350.08) | 1213.86 (379.24)
  Week 24: IgM (n=21,15,24,12,35,48,44,0,34,17,22) | 145.71 (86.21) | 144.73 (73.08) | 161.96 (62.54) | 153.08 (69.05) | 122.46 (46.08) | 140.06 (59.51) | 128.25 (56.26) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 143.29 (73.11) | 153.24 (80.78) | 167.95 (82.86)
  Week 24: IgA (n=21,15,24,12,35,48,43,0,34,17,22) | 305.62 (160.91) | 435.00 (405.07) | 237.00 (87.21) | 287.50 (107.94) | 294.97 (136.28) | 280.65 (118.50) | 232.51 (100.39) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 294.35 (131.76) | 329.65 (152.74) | 305.18 (150.23)

33. Other Pre Specified Outcome: Change From Baseline in Serum Immunoglobulin G (IgG), Immunoglobulin M (IgM) and Immunoglobulin A (IgA) Levels at Week 24
Description: Blood samples for immunoglobulin assessments were obtained to determine change from baseline in serum IgG, IgM, and IgA levels.
Time Frame: Baseline, Week 24/ ET
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline measure. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 18 | 15 | 22 | 11 | 32 | 46 | 41 | 32 | 15 | 20
mg/dL
  IgG | -13.50 (159.02) | -114.27 (321.37) | -71.55 (152.89) | -145.36 (267.20) | -53.81 (164.31) | -131.50 (183.76) | -86.44 (175.79) | -49.81 (192.28) | 31.00 (129.17) | -59.75 (163.33)
  IgM | 7.83 (21.88) | -9.73 (35.26) | -11.86 (25.02) | -3.73 (27.32) | 4.25 (16.41) | -17.02 (41.65) | -22.73 (33.64) | -3.69 (46.72) | 3.00 (30.44) | -2.50 (37.27)
  IgA | 6.28 (44.81) | 7.07 (164.76) | -38.50 (55.58) | -45.36 (59.51) | -24.53 (48.01) | -42.50 (72.55) | -68.41 (104.16) | -26.03 (82.04) | 8.60 (45.09) | -18.15 (52.51)

34. Other Pre Specified Outcome: Fluorescence Activated Cell Sorting (FACS) Lymphocyte Biomarkers
Description: The following biomarkers were assessed: Cluster of Differentiation 3 (CD3), CD4, CD8, CD19 and CD56. FACS analysis for lymphocyte subset markers were used to assess the effects of repeated doses of CP-690,550.
Time Frame: Baseline, Week 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cells per micro liter (cells/mcL)
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 30 | 6 | 35 | 7 | 29 | 37 | 34 | 32 | 19 | 40 | 12
cells per micro liter (cells/mcL)
  Baseline: CD3 (n=30,0,35,0,29,37,34,32,0,40,0) | 1.29 (0.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.31 (0.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.31 (0.73) | 1.24 (0.61) | 1.30 (0.51) | 1.36 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.17 (0.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: CD4 (n=30,0,35,0,29,37,34,32,0,40,0) | 0.84 (0.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.93 (0.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.93 (0.56) | 0.85 (0.49) | 0.89 (0.35) | 0.91 (0.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.80 (0.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: CD8 (n=30,0,35,0,29,37,34,32,0,40,0) | 0.44 (0.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.37 (0.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.37 (0.26) | 0.37 (0.19) | 0.40 (0.21) | 0.43 (0.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.35 (0.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: CD19 (n=30,0,34,0,29,37,34,32,0,40,0) | 0.21 (0.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.20 (0.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.22 (0.23) | 0.19 (0.09) | 0.20 (0.12) | 0.18 (0.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.16 (0.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: CD56 (n=30,0,34,0,29,37,34,32,0,40,0) | 0.15 (0.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.14 (0.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.14 (0.10) | 0.14 (0.12) | 0.14 (0.10) | 0.14 (0.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.12 (0.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: CD3 (n=16,6,17,7,22,29,26,0,19,9,12) | 1.16 (0.67) | 1.45 (0.57) | 1.45 (0.82) | 1.20 (0.46) | 1.10 (0.43) | 1.27 (0.61) | 1.14 (0.36) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 1.46 (0.48) | 1.63 (0.69) | 1.26 (0.57)
  Week 24: CD4 (n=16,6,17,7,22,29,26,0,19,9,12) | 0.75 (0.42) | 0.87 (0.33) | 1.01 (0.65) | 0.86 (0.35) | 0.77 (0.30) | 0.92 (0.51) | 0.82 (0.26) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.98 (0.35) | 1.01 (0.52) | 0.91 (0.45)
  Week 24: CD8 (n=16,6,17,7,22,29,26,0,19,9,12) | 0.38 (0.26) | 0.58 (0.43) | 0.42 (0.25) | 0.30 (0.13) | 0.31 (0.18) | 0.33 (0.15) | 0.32 (0.14) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.45 (0.34) | 0.58 (0.34) | 0.33 (0.14)
  Week 24: CD19 (n=16,6,17,7,22,29,25,0,19,9,12) | 0.23 (0.18) | 0.27 (0.14) | 0.22 (0.11) | 0.27 (0.15) | 0.17 (0.11) | 0.31 (0.16) | 0.24 (0.09) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.29 (0.15) | 0.12 (0.05) | 0.31 (0.21)
  Week 24: CD56 (n=16,6,17,7,22,29,26,0,19,9,12) | 0.10 (0.06) | 0.12 (0.09) | 0.11 (0.08) | 0.08 (0.10) | 0.07 (0.05) | 0.05 (0.05) | 0.04 (0.03) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.09 (0.09) | 0.15 (0.12) | 0.07 (0.06)

35. Other Pre Specified Outcome: Change From Baseline in Fluorescence Activated Cell Sorting (FACS) Lymphocyte Biomarkers at Week 24
Description: The following biomarkers were assessed: CD3, CD4, CD8, CD19 and CD56. FACS analysis for lymphocyte subset markers were used to assess the effects of repeated doses of CP-690,550.
Time Frame: Baseline, Week 24/ ET
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 9 | 5 | 11 | 7 | 18 | 21 | 20 | 17 | 7 | 11
cells/mcL
  CD3 | 0.01 (0.77) | 0.00 (0.44) | 0.07 (0.62) | 0.07 (0.39) | -0.19 (0.52) | 0.01 (0.45) | -0.13 (0.44) | 0.12 (0.60) | 0.36 (0.38) | 0.20 (0.50)
  CD4 | -0.03 (0.50) | -0.05 (0.31) | 0.06 (0.48) | 0.07 (0.30) | -0.16 (0.41) | 0.03 (0.32) | -0.11 (0.31) | 0.08 (0.49) | 0.20 (0.33) | 0.18 (0.37)
  CD8 | 0.01 (0.28) | 0.04 (0.14) | 0.01 (0.17) | -0.01 (0.14) | -0.03 (0.18) | -0.02 (0.15) | -0.03 (0.14) | 0.04 (0.19) | 0.11 (0.11) | 0.03 (0.14)
  CD19 | 0.03 (0.24) | 0.01 (0.10) | -0.00 (0.17) | 0.07 (0.07) | -0.03 (0.21) | 0.12 (0.14) | 0.06 (0.10) | 0.09 (0.13) | 0.02 (0.03) | 0.13 (0.12)
  CD56 | -0.05 (0.05) | 0.03 (0.08) | -0.03 (0.05) | -0.06 (0.15) | -0.06 (0.09) | -0.06 (0.07) | -0.08 (0.04) | -0.03 (0.08) | 0.01 (0.07) | -0.05 (0.08)

36. Other Pre Specified Outcome: Medical Outcome Study- Sleep Scale (MOS-SS)
Description: Participant-rated questionnaire to assess key constructs of sleep over the past week. Consists of a 12-item based on 7 sub scales: sleep disturbance (SD), snoring (Sno), awakened short of breath (ASOB) or with headache, sleep adequacy (Ade), and somnolence (Som) (range:0-100); sleep quantity (Qua)(range:0-24), and optimal (Opt) sleep (yes: 1, no: 0)and nine item index measures of sleep disturbance were constructed to provide composite scores: sleep problem summary (SPS) and overall sleep problems (OSP). Except sleep adequacy, optimal sleep and quantity, higher scores=greater impairment. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 2, 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 15 | 51 | 15 | 49 | 61 | 57 | 53 | 40 | 59 | 24
units on a scale
  Baseline: SPS (n=54,0,51,0,49,61,57,53,0,58,0) | 45.06 (22.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.56 (19.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.86 (17.35) | 44.86 (17.60) | 44.39 (23.35) | 44.72 (22.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.77 (18.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: OSP (n=54,0,51,0,49,61,57,53,0,58,0) | 44.87 (22.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 48.34 (19.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.51 (18.35) | 45.82 (15.79) | 45.77 (22.68) | 45.94 (22.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.12 (18.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Ade (n=54,0,51,0,49,61,57,53,0,58,0) | 40.74 (27.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.31 (27.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.10 (23.73) | 41.31 (24.93) | 40.18 (27.87) | 39.81 (27.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.62 (23.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: A SOB (n=54,0,51,0,49,61,57,53,0,58,0) | 22.96 (22.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.41 (30.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.82 (22.35) | 23.61 (27.69) | 27.72 (30.18) | 21.51 (28.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 23.10 (27.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: SD (n=54,0,51,0,49,61,57,53,0,58,0) | 46.60 (28.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 52.40 (25.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.52 (25.73) | 48.34 (22.61) | 45.09 (28.53) | 47.90 (28.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.72 (24.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Opt (n=54,0,51,0,49,61,57,53,0,59,0) | 0.31 (0.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.45 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.51 (0.51) | 0.31 (0.47) | 0.42 (0.50) | 0.57 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.47 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Qua (n=54,0,51,0,49,61,57,53,0,59,0) | 6.11 (1.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.51 (1.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.76 (1.39) | 6.59 (1.76) | 6.33 (1.38) | 6.72 (2.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.63 (1.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Sno (n=54,0,51,0,49,61,57,53,0,58,0) | 30.00 (34.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.39 (36.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.84 (34.14) | 33.11 (31.60) | 32.28 (32.02) | 42.26 (32.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.24 (31.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Som (n=54,0,51,0,49,61,57,53,0,58,0) | 36.05 (22.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.69 (21.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.05 (22.27) | 38.91 (25.57) | 38.36 (18.78) | 38.74 (25.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.68 (21.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SPS (n=54,0,50,0,48,59,57,52,0,56,0) | 41.79 (21.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.73 (19.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.22 (17.41) | 37.57 (17.68) | 35.50 (21.27) | 38.46 (21.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.18 (19.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: OSP (n=54,0,50,0,48,59,57,52,0,56,0) | 41.64 (20.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.19 (19.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.61 (17.17) | 37.75 (16.80) | 36.15 (21.04) | 39.24 (21.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.35 (18.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Ade (n=54,0,51,0,48,59,57,52,0,56,0) | 46.11 (27.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.14 (26.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.04 (25.54) | 47.80 (26.40) | 52.63 (29.00) | 48.65 (30.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.21 (25.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: A SOB (n=54,0,50,0,48,59,57,52,0,56,0) | 23.33 (24.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.80 (28.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.25 (28.03) | 19.32 (23.18) | 23.16 (28.98) | 19.23 (25.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.79 (22.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SD (n=54,0,50,0,48,59,57,52,0,56,0) | 42.01 (25.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.48 (25.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.81 (23.40) | 38.24 (23.34) | 36.69 (26.47) | 39.16 (27.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.32 (24.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Opt (n=54,0,51,0,48,60,57,53,0,58,0) | 0.39 (0.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.35 (0.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.60 (0.49) | 0.45 (0.50) | 0.47 (0.50) | 0.43 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.48 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Qua (n=54,0,51,0,48,60,57,52,0,57,0) | 6.31 (1.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.41 (1.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.98 (1.23) | 6.85 (1.69) | 6.72 (1.26) | 6.71 (2.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.74 (1.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Sno (n=54,0,51,0,48,59,57,52,0,56,0) | 27.04 (28.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.16 (30.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.83 (30.02) | 30.85 (29.79) | 32.28 (28.97) | 40.38 (31.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.43 (29.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Som (n=54,0,51,0,48,59,57,52,0,56,0) | 36.05 (21.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.20 (18.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.69 (22.20) | 31.75 (22.57) | 30.53 (18.17) | 38.33 (28.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.86 (21.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SPS (n=44,0,46,0,45,57,53,45,0,45,0) | 35.61 (22.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.48 (21.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.85 (16.91) | 35.09 (18.32) | 31.26 (22.84) | 36.37 (20.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.56 (18.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: OSP (n=44,0,46,0,45,57,53,45,0,45,0) | 36.44 (22.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.93 (21.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.51 (17.81) | 35.19 (17.56) | 32.11 (22.33) | 37.09 (20.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.26 (18.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ade (n=44,0,46,0,45,57,53,45,0,45,0) | 58.18 (27.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.30 (28.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 48.67 (24.36) | 49.82 (28.06) | 57.55 (31.06) | 49.56 (24.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 53.11 (24.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: A SOB (n=44,0,46,0,45,57,53,45,0,45,0) | 19.09 (21.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.17 (26.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.00 (22.40) | 17.19 (19.80) | 23.02 (27.00) | 19.11 (24.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.44 (23.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SD (n=44,0,46,0,45,57,53,45,0,45,0) | 38.58 (27.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.39 (26.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.94 (25.31) | 36.47 (25.90) | 31.30 (25.45) | 37.22 (28.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.08 (21.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Opt (n=44,0,46,0,45,57,54,45,0,46,0) | 0.45 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.43 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.47 (0.50) | 0.51 (0.50) | 0.52 (0.50) | 0.58 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.61 (0.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Qua (n=44,0,46,0,45,56,53,45,0,46,0) | 6.77 (1.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.65 (1.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.91 (1.28) | 6.80 (1.55) | 6.68 (1.25) | 6.78 (1.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.09 (1.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Sno (n=44,0,46,0,45,57,53,45,0,45,0) | 30.45 (30.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.96 (33.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.67 (32.59) | 30.53 (25.10) | 28.68 (29.49) | 36.89 (32.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 23.56 (25.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Som (n=44,0,46,0,45,57,53,45,0,45,0) | 34.70 (22.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.59 (21.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.19 (24.39) | 29.12 (21.44) | 27.80 (19.42) | 35.26 (26.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.37 (19.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: SPS (n=24,15,29,15,43,55,52,0,40,20,24) | 30.83 (18.55) | 45.56 (20.77) | 32.07 (18.22) | 39.33 (22.54) | 33.72 (18.42) | 34.18 (18.66) | 33.85 (21.69) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 32.75 (19.48) | 31.17 (21.20) | 33.19 (17.54)
  Week 24: OSP (n=24,15,29,15,43,55,52,0,40,20,24) | 30.93 (18.06) | 43.37 (19.86) | 32.32 (18.93) | 39.67 (21.03) | 34.30 (18.69) | 34.18 (17.79) | 33.57 (19.91) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 33.14 (19.80) | 31.39 (19.85) | 33.89 (15.61)
  Week 24: Ade (n=24,15,29,15,43,55,52,0,40,20,24) | 60.00 (28.89) | 40.67 (29.39) | 59.66 (26.52) | 45.33 (26.96) | 53.26 (24.08) | 50.00 (28.41) | 51.73 (30.53) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 59.50 (25.31) | 60.50 (25.64) | 54.58 (22.06)
  Week 24: A SOB (n=24,15,29,15,43,55,52,0,40,20,24) | 25.00 (27.82) | 36.00 (21.65) | 24.14 (27.97) | 30.67 (33.69) | 22.79 (29.79) | 21.45 (21.72) | 23.46 (26.78) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 25.50 (30.38) | 17.00 (23.64) | 13.33 (18.34)
  Week 24: SD (n=24,15,29,15,43,55,52,0,40,20,24) | 29.79 (21.33) | 41.58 (23.29) | 34.27 (24.80) | 38.58 (24.30) | 33.58 (22.98) | 33.09 (23.23) | 31.59 (23.31) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 33.81 (27.14) | 33.13 (24.58) | 36.46 (21.42)
  Week 24: Opt (n=24,15,29,15,43,55,52,0,40,20,24) | 0.58 (0.50) | 0.31 (0.48) | 0.55 (0.51) | 0.33 (0.49) | 0.72 (0.45) | 0.38 (0.49) | 0.50 (0.50) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.55 (0.50) | 0.75 (0.44) | 0.50 (0.51)
  Week 24: Qua (n=24,14,29,15,43,55,52,0,40,20,24) | 7.04 (1.63) | 7.00 (1.41) | 6.83 (1.42) | 6.60 (1.35) | 7.14 (1.06) | 6.73 (1.60) | 6.92 (1.44) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 6.95 (1.41) | 7.20 (1.06) | 7.00 (1.25)
  Week 24: Sno (n=24,15,29,15,43,55,52,0,40,20,24) | 23.33 (20.14) | 33.33 (36.77) | 38.62 (32.04) | 36.00 (33.97) | 34.42 (31.27) | 28.73 (27.96) | 31.54 (29.73) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 40.50 (32.18) | 34.00 (31.19) | 32.50 (24.18)
  Week 24: Som (n=24,15,29,15,43,55,52,0,40,20,24) | 29.44 (20.80) | 30.67 (18.14) | 26.44 (19.48) | 31.11 (22.21) | 30.39 (17.54) | 27.39 (20.47) | 26.54 (17.83) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 30.17 (22.80) | 28.00 (18.17) | 28.33 (17.72)

37. Other Pre Specified Outcome: Change From Baseline in Medical Outcome Study- Sleep Scale (MOS-SS) at Week 2, 12 and 24/ET
Description: Participant-rated questionnaire to assess key constructs of sleep over the past week. Consists of a 12-item based on 7 subscales: sleep disturbance (SD), snoring (Sno), awakened short of breath (A SOB) or with headache, sleep adequacy (Ade), and somnolence (Som) (range: 0-100); sleep quantity (Qua) (range: 0-24), and optimal (Opt) sleep (yes: 1, no: 0) and 9 item index measures of sleep disturbance were constructed to provide 2 composite scores: sleep problem summary (SPS) and overall sleep problems (OSP). Except sleep adequacy, optimal sleep and quantity, higher scores=greater impairment. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range*100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 2, 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 16 | 51 | 15 | 48 | 60 | 57 | 53 | 40 | 58 | 24
units on a scale
  Week 2: SPS (n=54,0,50,0,48,59,57,52,0,55,0) | -3.27 (14.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.13 (12.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.50 (18.09) | -7.12 (15.14) | -8.89 (17.59) | -6.99 (16.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.85 (15.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: OSP (n=54,0,50,0,48,59,57,52,0,55,0) | -3.23 (13.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.36 (11.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.62 (17.59) | -7.95 (15.26) | -9.62 (16.95) | -7.41 (15.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.89 (16.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Ade (n=54,0,51,0,48,59,57,52,0,55,0) | 5.37 (20.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.18 (20.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.83 (23.95) | 7.29 (23.33) | 12.46 (25.44) | 10.00 (24.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.82 (19.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: A SOB (n=54,0,50,0,48,59,57,52,0,55,0) | 0.37 (21.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.20 (26.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.83 (25.75) | -4.07 (30.80) | -4.56 (21.39) | -1.92 (23.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.18 (18.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SD (n=54,0,50,0,48,59,57,52,0,55,0) | -4.58 (18.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.25 (14.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.38 (22.80) | -9.83 (19.04) | -8.40 (23.32) | -9.66 (18.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.89 (23.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Opt (n=54,0,51,0,48,60,57,53,0,58,0) | 0.07 (0.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.10 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.08 (0.50) | 0.13 (0.50) | 0.05 (0.61) | -0.13 (0.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 (0.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Qua (n=54,0,51,0,48,60,57,52,0,57,0) | 0.20 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.10 (1.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.19 (1.16) | 0.20 (1.22) | 0.39 (1.06) | 0.02 (1.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.11 (1.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Sno (n=54,0,51,0,48,59,57,52,0,55,0) | -2.96 (19.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.24 (22.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.67 (15.34) | -1.69 (19.75) | 0.00 (27.26) | -1.15 (16.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.36 (18.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Som (n=54,0,51,0,48,59,57,52,0,55,0) | -0.00 (19.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.49 (17.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.14 (18.63) | -6.33 (19.20) | -7.84 (17.05) | -0.90 (16.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.21 (14.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SPS (n=44,0,46,0,45,57,53,45,0,44,0) | -8.56 (19.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.59 (17.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.74 (17.05) | -9.82 (18.09) | -11.70 (18.44) | -6.96 (16.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.32 (18.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: OSP (n=44,0,46,0,45,57,53,45,0,44,0) | -7.16 (18.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.85 (16.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.73 (16.87) | -10.75 (17.25) | -12.16 (17.51) | -7.36 (15.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.19 (18.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ade (n=44,0,46,0,45,57,53,45,0,44,0) | 15.45 (28.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.52 (26.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.56 (25.33) | 9.30 (27.38) | 15.28 (26.79) | 9.33 (27.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.14 (21.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: A SOB (n=44,0,46,0,45,57,53,45,0,44,0) | -6.36 (19.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.83 (31.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.89 (20.96) | -6.67 (25.45) | -3.40 (24.72) | -0.89 (27.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.82 (23.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SD (n=44,0,46,0,45,57,53,45,0,44,0) | -6.56 (21.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.24 (22.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.89 (25.34) | -12.52 (22.44) | -12.08 (23.49) | -9.11 (21.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.04 (25.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Opt (n=44,0,46,0,45,57,54,45,0,46,0) | 0.09 (0.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.02 (0.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.02 (0.54) | 0.19 (0.52) | 0.07 (0.64) | -0.04 (0.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.11 (0.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Qua (n=44,0,46,0,45,56,53,45,0,46,0) | 0.52 (1.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.15 (1.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.16 (1.11) | 0.27 (1.36) | 0.30 (1.34) | 0.07 (2.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.35 (1.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Sno (n=44,0,46,0,45,57,53,45,0,44,0) | 1.82 (29.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.91 (28.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.78 (20.37) | -1.40 (25.60) | -1.51 (19.55) | -3.11 (25.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.36 (23.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Som (n=44,0,46,0,45,57,53,45,0,44,0) | 0.30 (22.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.96 (17.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.41 (21.63) | -8.30 (22.37) | -9.43 (18.65) | -1.04 (21.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.67 (18.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: SPS (n=24,15,29,15,43,55,52,0,40,19,24) | -8.89 (16.32) | -11.78 (25.66) | -12.18 (17.21) | -5.11 (21.34) | -6.90 (18.39) | -11.09 (18.31) | -10.00 (20.69) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -11.50 (22.93) | -8.60 (13.21) | -11.94 (22.76)
  Week 24: OSP (n=24,15,29,15,43,55,52,0,40,19,24) | -8.43 (14.30) | -12.48 (24.26) | -14.44 (17.70) | -8.52 (19.53) | -9.10 (18.33) | -12.14 (17.76) | -11.68 (17.94) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -12.25 (20.59) | -10.35 (13.71) | -12.64 (19.16)
  Week 24: Ade (n=24,15,29,15,43,55,52,0,40,19,24) | 12.92 (30.29) | 11.33 (32.04) | 9.66 (26.39) | 4.67 (27.74) | 7.21 (26.76) | 10.00 (29.19) | 10.77 (26.33) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 21.00 (26.68) | 13.16 (16.68) | 17.50 (28.93)
  Week 24: A SOB (n=24,15,29,15,43,55,52,0,40,19,24) | 4.17 (25.01) | 1.33 (34.20) | -8.97 (32.33) | 6.67 (31.77) | 0.93 (27.59) | -2.91 (27.60) | -3.08 (29.48) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 5.00 (29.26) | -5.26 (16.11) | -5.83 (27.96)
  Week 24: SD (n=24,15,29,15,43,55,52,0,40,19,24) | -11.88 (20.92) | -16.42 (30.92) | -16.98 (24.82) | -11.50 (23.66) | -12.33 (24.35) | -16.14 (22.21) | -13.20 (23.25) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -13.44 (26.54) | -10.92 (20.62) | -16.15 (23.75)
  Week 24: Opt (n=24,16,29,15,43,55,52,0,40,20,24) | 0.17 (0.56) | 0.00 (0.52) | 0.07 (0.53) | -0.13 (0.64) | 0.23 (0.53) | 0.05 (0.52) | 0.08 (0.52) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -0.08 (0.62) | 0.20 (0.62) | 0.08 (0.50)
  Week 24: Qua (n=24,14,29,15,43,55,52,0,40,20,24) | 0.83 (0.92) | 0.57 (1.02) | 0.45 (1.50) | -0.27 (1.53) | 0.37 (1.20) | 0.18 (1.59) | 0.62 (1.24) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 0.23 (2.39) | 0.50 (1.19) | 0.33 (1.31)
  Week 24: Sno (n=24,15,29,15,43,55,52,0,40,19,24) | 0.00 (26.38) | -4.00 (18.82) | -4.83 (27.60) | -2.67 (19.81) | 2.33 (26.26) | -2.18 (24.55) | 0.77 (27.99) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 2.50 (22.27) | -2.11 (39.38) | 5.83 (18.16)
  Week 24: Som (n=24,15,29,15,43,55,52,0,40,19,24) | 0.00 (19.66) | -13.33 (20.00) | -11.95 (21.04) | -9.78 (19.33) | -7.29 (18.56) | -10.42 (23.40) | -11.03 (22.05) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | -5.50 (23.24) | -5.26 (16.27) | -2.50 (13.59)

38. Other Pre Specified Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-Fatigue is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 2, 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 15 | 51 | 15 | 49 | 60 | 57 | 53 | 40 | 59 | 24
units on a scale
  Baseline (n=54,0,51,0,49,60,57,53,0,59,0) | 28.39 (11.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.90 (9.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.84 (11.85) | 26.75 (12.19) | 25.74 (11.32) | 25.87 (11.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.49 (9.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=54,0,51,0,48,60,56,52,0,57,0) | 29.06 (10.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.52 (9.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.31 (11.84) | 31.80 (11.57) | 31.66 (10.99) | 29.15 (12.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.23 (10.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,45,56,54,45,0,46,0) | 34.57 (10.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.37 (10.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.11 (11.29) | 37.11 (11.50) | 35.30 (11.63) | 30.58 (10.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.09 (10.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=24,15,29,15,43,55,52,0,40,20,24) | 35.21 (12.24) | 31.53 (9.98) | 37.48 (10.08) | 31.80 (8.79) | 35.00 (10.34) | 35.82 (11.59) | 34.03 (10.87) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 34.90 (10.47) | 35.45 (7.27) | 37.25 (8.52)

39. Other Pre Specified Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Week 2, 12 and 24/ET
Description: as for outcome 38
Time Frame: Baseline, Week 2, 12, 24/ ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 54 | 15 | 51 | 15 | 48 | 59 | 56 | 52 | 40 | 57 | 24
units on a scale
  Week 2 (n=54,0,51,0,48,59,56,52,0,57,0) | 0.67 (7.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.62 (7.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.38 (9.76) | 5.10 (9.32) | 6.07 (10.34) | 3.54 (9.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.70 (8.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=44,0,46,0,45,55,54,45,0,46,0) | 5.14 (9.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.00 (8.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.47 (8.70) | 9.40 (11.52) | 8.85 (11.84) | 3.78 (11.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.33 (9.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=24,15,29,15,43,55,52,0,40,20,24) | 4.96 (10.75) | 5.93 (9.93) | 6.97 (8.97) | 9.13 (6.83) | 8.81 (8.86) | 8.73 (11.87) | 7.59 (9.93) | NA (NA) — Data not available as all adalimumab participants received CP-690,550 5 mg after Week 12. | 7.80 (12.39) | 8.90 (8.72) | 8.63 (6.01)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Adalimumab | Adalimumab to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/17 | 1/34 | 0/17 | 0/49 | 1/61 | 4/57 | 0/9 | 4/44 | 2/34 | 0/25
Other Adverse Events (participants affected / at risk) | 18/37 | 5/17 | 18/34 | 6/17 | 27/49 | 31/61 | 31/57 | 5/9 | 26/44 | 14/34 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=37) | CP-690,550 1 mg to CP-690,550 5 mg (R) (N=17) | CP-690,550 3 mg (N=34) | CP-690,550 3 mg to CP-690,550 5 mg (R) (N=17) | CP-690,550 5 mg (N=49) | CP-690,550 10 mg (N=61) | CP-690,550 15 mg (N=57) | Adalimumab (N=9) | Adalimumab to CP-690,550 5 mg (R) (N=44) | Placebo (N=34) | Placebo to CP-690,550 5 mg (R) (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CP-690,550 1 mg (N=37) | CP-690,550 1 mg to CP-690,550 5 mg (R) (N=17) | CP-690,550 3 mg (N=34) | CP-690,550 3 mg to CP-690,550 5 mg (R) (N=17) | CP-690,550 5 mg (N=49) | CP-690,550 10 mg (N=61) | CP-690,550 15 mg (N=57) | Adalimumab (N=9) | Adalimumab to CP-690,550 5 mg (R) (N=44) | Placebo (N=34) | Placebo to CP-690,550 5 mg (R) (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3 | 0 | 3 | 4 | 1 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 2 | 3 | 2 | 0 | 2 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 1 | 2 | 2 | 4 | 0 | 3 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 0 | 1 | 1 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 2 | 1 | 5 | 3 | 6 | 0 | 2 | 2 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram RR interval prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 6 | 3 | 0 | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0/1 | 1 | 0 | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 1
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.